### The GlaxoSmithKline group of companies

208470

| Division | : Worldwide Development |
|------------------|-------------------------------------|
| Information Type | : Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for Open-Label Pilot Study to Assess the Safety, Tolerability and Antitumor Activity of Genetically Engineered NY-ESO-1 Specific (c259) T-cells Alone or in Combination with Pembrolizumab in HLA-A2+ Subjects with NY-ESO-1 and/or LAGE-1a Positive Relapsed and Refractory Multiple Myeloma |
|---|---|---|
| <b>Compound Number</b> | : | GSK3377794 |
| <b>Effective Date</b> | : | 23-APR-2021 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the abbreviated Clinical Study Report for Protocol 208470.
- This RAP is intended to describe the planned safety, tolerability and efficacy analyses required for the study.
- This RAP will be provided to study team members to convey the planned content of the Statistical Analysis Complete (SAC) deliverable.

# **RAP Author(s):**

| R-2021 |
|--------|
| - |

Copyright 2021 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

208470

# **RAP Team Reviewer (Method: Email):**

| Approver | Date |
|---|---|
| PPD | 29-MAR-2021 |
| Statistician (Contingent Worker),<br>GlaxoSmithKline | |
| PPD | 29-MAR-2021 |
| Principal Programmer (Oncology Clinical Programming), GlaxoSmithKline | |
| PPD | 31-MAR-2021 |
| Principal Statistical Programmer,<br>PAREXEL | |
| PPD | 31-MAR-2021 |
| Clinical Scientist (Oncology Clinical Development), GlaxoSmithKline | |
| PPD | 08-APR-2021 |
| Quantitative Clinical Pharmacology<br>Director (Oncology CPMS),<br>GlaxoSmithKline | |
| PPD | 06-APR-2021 |
| Clinical Biomarker Lead (Oncology Cell | |
| Therapy, EMU), GlaxoSmithKline | |

# **Clinical Statistics and Clinical Programming Line Approvals (Method: Email):**

| Approver | Date |
|---|---|
| PPD | 23-APR-2021 |
| Statistics, Director, Oncology Clinical<br>Statistics, GlaxoSmithKline | |
| PPD | 22-APR-2021 |
| Director, Oncology Clinical<br>Programming, GlaxoSmithKline | |

208470

# **TABLE OF CONTENTS**

| | | PAGE |
|---|---|---|
| 1. | INTRODUCTION | 7 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | q |
| | 2.1. Change to Protocol Specified Statistical Analysis Plan | |
| | 2.2. Study Objective(s) and Endpoint(s) | |
| | 2.3. Study Design | |
| | 2.4. Statistical Analyses | |
| | • | |
| 3. | PLANNED ANALYSES | |
| | 3.1. Safety Monitoring Review for TLTs | |
| | 3.1.1. Predictive Probabilities | |
| | 3.2. Interim Analyses | |
| | 3.3. Final Analysis | 18 |
| 4. | ANALYSIS POPULATIONS | 19 |
| | 4.1. Protocol Deviations | |
| 5. | CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | 00 |
| | CONVENTIONS | |
| | 5.1. Study Treatment & Sub-group Display Descriptors | |
| | 5.2. Baseline Definitions | |
| | 5.3. Multicentre Studies | |
| | 5.4. Examination of Covariates, Other Strata and Subgroups | |
| | <ul><li>5.5. Multiple Comparisons and Multiplicity</li><li>5.6. Other Considerations for Data Analyses and Data Handling</li></ul> | 21 |
| | Conventions | 21 |
| 6. | STUDY POPULATION ANALYSES | |
| | 6.1. Overview of Planned Study Population Analyses | |
| | 6.2. Disposition of Participants | |
| | 6.3. Protocol Deviations | |
| | 6.4. Demographic and Baseline Characteristics | |
| | 6.5. Prior and Concomitant Medications | |
| | 6.6. Study Treatment Exposure | |
| | 6.7. Anti-Cancer Therapies | |
| | 6.7.1. Prior Anti-Cancer Therapies | |
| | 6.7.2. On-Study Anti-Cancer Therapies | 25 |
| 7. | EFFICACY ANALYSES | 27 |
| | 7.1. Primary Efficacy Analyses | |
| | 7.1.1. Primary Endpoint/Variable: Overall Response Rate (ORR) | |
| | 7.1.1.1. Best Overall Response | |
| | 7.1.1.2. Overall Response Rate | |
| | 7.1.1.3. Definition of Adequate Assessment | |
| | 7.1.1.4. Date Associated with Response | |
| | 7.1.1.5. Confirmed Response | |
| | 7.1.2. Summary Measurement | |
| | 7.1.3. Population of Interest | 30 |

| | | 7.1.4. | Strategy for Intercurrent Events | |
|---|---|---|---|---|
| | | 7.1.5. | Statistical Analyses / Methods | |
| | 7.2. | | ary Efficacy Analyses | |
| | | 7.2.1. | Endpoints/Variables | |
| | | | 7.2.1.1. Time to Response (TTR) | |
| | | | 7.2.1.2. Duration of Response (DoR) | |
| | | | 7.2.1.3. Progression Free Survival (PFS) | 33 |
| | | 7.2.2. | Summary Measure | 35 |
| | | | 7.2.2.1. Time to Response (TTR) | |
| | | | 7.2.2.2. Duration of Response | |
| | | | 7.2.2.3. Progression Free Survival | |
| | | 7.2.3. | Population of Interest | |
| | | 7.2.4. | Statistical Analyses / Methods | |
| | 7.3. | | ory Efficacy Analyses | |
| | | 7.3.1. | Endpoints/Variables | |
| | | <b>7</b> 0 0 | 7.3.1.1. Overall Survival (OS) | |
| | | 7.3.2. | Summary Measure | |
| | | 7.3.3. | Population of Interest | |
| | | 7.3.4. | Statistical Analyses / Methods | 36 |
| 0 | CAFE | T\/ | VOEC | 20 |
| 8. | | | YSES | |
| | 8.1. | | Events Analyses | |
| | 8.2. | | Events of Special Interest (AESI) Analyses | 40 |
| | | 8.2.1. | Cytokine Release Syndrome (CRS) and Graft versus Host Disease (GvHD) | 11 |
| | 8.3. | Clinical | | |
| | 0.3. | 8.3.1. | Laboratory Analyses | |
| | 8.4. | | Analyses of Liver Function Tests (LFT)afety Analyses | |
| | 0.4. | 8.4.1. | Performance Status | |
| | | 8.4.2. | ECG | |
| | | 8.4.3. | Pregnancies | |
| | | 8.4.4. | Vital Signs | |
| | | 8.4.5. | Replication Competent Lentivirus (RCL) and Persistence | 43 |
| | | 0.4.5. | of NY-ESO-1 <sup>c259</sup> T | 46 |
| | | 8.4.6. | COVID-19 | |
| | | 0.4.0. | OOVID-19 | |
| 9. | PHAR | MACOKI | NETIC ANALYSES | 46 |
| ٥. | 9.1. | | Pharmacokinetic Analyses | |
| | 0.1. | 9.1.1. | Endpoint / Variables | 46 |
| | | 0.1.1. | 9.1.1.1. Drug Concentration Measures | |
| | | | 9.1.1.2. Derived Pharmacokinetic Parameters | |
| | | 9.1.2. | Summary Measure | |
| | | 9.1.3. | Population of Interest | |
| | | 0.1.0. | | |
| 10. | BIOM | ARKER A | NALYSES | 49 |
| | 10.1. | | er Analyses | |
| | | 10.1.1. | · | |
| | | 10.1.2. | | |
| | | | 10.1.2.1. Anti-NYESO-1 Antibody Formation | |
| | | 10.1.3. | Population of Interest | |
| | | 10.1.4. | Statistical Analyses / Methods | |
| | | | • | _ |

208470

| 11. | POPUI | _ATION P | HARMACOKINETIC (POPPK) ANALYSES | .49 |
|---|---|---|---|---|
| 12. | PHAR | MACOKIN | ETIC / PHARMACODYNAMIC ANALYSES | .49 |
| 13. | REFER | RENCES | | . 50 |
| 14 | ΔPPFN | IDICES | | 51 |
| | 14.1. | <b>Appendix</b> | 1: Protocol Deviation Management and Definitions for Per | |
| | 14.2. | | Population2: Schedule of Activities | |
| | 14.2. | | Protocol Defined Schedule of Events | |
| | | | Schedule of Procedures in Long-Term Follow-up prior to | . 52 |
| | | 17.2.2. | Transfer to LTFU Protocol | 59 |
| | 14.3. | Annendix | 3: Assessment Windows | |
| | | | Definitions of Assessment Windows for Analyses | |
| | 14.4. | | 4: Study Phases and Treatment Emergent Adverse | |
| | | | | .62 |
| | | | Study Phase | |
| | | | 14.4.1.1. Study Phases for Concomitant Medication | .62 |
| | | | 14.4.1.2. Study Phases for Anti-Cancer Therapy/Surgery | |
| | | | Treatment Emergent Flag for Adverse Events | |
| | 14.5. | | 5: Data Display Standards & Handling Conventions | |
| | | 14.5.1. | Reporting Process | |
| | | 14.5.2. | Reporting Standards | |
| | 44.0 | 14.5.3. | Reporting Standards for Pharmacokinetic Data | |
| | 14.6. | Appendix 14.6.1. | 6: Derived and Transformed Data | |
| | | 14.6.1. | GeneralStudy Population | |
| | | 14.6.2. | Safety | |
| | | | Efficacy | |
| | 14.7. | | 7: Reporting Standards for Missing Data | |
| | | | Premature Withdrawals | |
| | | | Handling of Missing Data | |
| | | | 14.7.2.1. Handling of Missing and Partial Dates | |
| | 14.8. | <b>Appendix</b> | 8: Values of Potential Clinical Importance | |
| | | 14.8.1. | Laboratory Values | .71 |
| | | | ECG | |
| | | | Vital Signs | |
| | 14.9. | | 9: Population Pharmacokinetic (PopPK) Analyses | |
| | | | 10: Pharmacokinetic / Pharmacodynamic Analyses | |
| | 14.11. | Appendix | 11: Abbreviations & Trademarks | .75 |
| | | | Abbreviations | |
| | 1110 | | Trademarks | |
| | 14.12. | | 12: List of Data Displays Data Display Numbering | |
| | | | Mock Example Shell Referencing | |
| | | | Deliverables | |
| | | | Study Population Tables | |
| | | | Efficacy Tables | |
| | | | Efficacy Figures | |
| | | | Safety Tables | |

# l Statistical Analysis Plan RAP 23 Apr 2021 | TMF-13337917 | 1.0

# CONFIDENTIAL

| | | 208470 |
|--------|----------------------------------------------------|--------|
| | 14.12.8. Safety Figures | 108 |
| | 14.12.9. Biomarkers Tables | |
| | 14.12.10. Pharmacokinetic Tables | 113 |
| | 14.12.11. Pharmacokinetic Figures | 114 |
| | 14.12.12.ICH Listings | 115 |
| | 14.12.13. Non-ICH Listings | 126 |
| 14.13. | Appendix 13: Example Mock Shells for Data Displays | 131 |
| 14.14. | Appendix 14: Combined Preferred Terms | 132 |
| | Appendix 15: Adverse Event Collapsing Rules | |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 208470:

| Protocol Revision Chronology: | | |
|---|---|---|
| Version 01 | 19-Dec-2016 | Original |
| Version 02<br>(Amendment 1) | 13-Mar-2017 | Changes included: - Integration of the sequential screening tests for HLA-genotyping and NY-ESO-1/LAGE-1a antigen expression level determination by RT-PCR Update to Pembrolizumab background Miscellaneous minor corrections/clarifications. |
| Version 03<br>(Amendment 2) | 24-Jul-2018 | Subsequent to the licensing of Adaptimmune product NY-ESO by GlaxoSmithKline (GSK), the purpose of this protocol amendment was to: - Delete or replace references to Adaptimmune or its staff with that of GSK and its authorized agents to align with the change of sponsorship. - Make administrative changes to align with GSK processes and procedures. - Make changes to lymphodepletion regimen. |
| Version 04<br>(Amendment 3) | 17-Oct-2018 | Changes made to the protocol were requested by the FDA as a result of safety events which included 2 reports of Guillain-Barré Syndrome in subjects who received chemotherapy and GSK3377794 during clinical trials. |
| Version 05<br>(Amendment 4) | 19-Sep-2019 | Several changes were made related to FDA requests, including updating Inclusion Criterion #5, adding study stopping rules, and updating Encephalopathy (now Immune Effector Cell-Associated Neurotoxicity or ICANS) and CRS grading and management criteria based upon American Society for Transplantation and Cellular Therapy, Lee, 2019 guidance. Also, changes were made to the lymphodepletion regimen for older subjects, and the randomization scheme was removed to first enrol subjects into Arm 1 (NY-ESO-1c259 T single infusion). |
| Version 06<br>(Amendment 5) | 24-Feb-2020 | This amendment restructured the protocol for a clearer presentation of the 3-part study design. The amendment also introduced the intent to enrol, treat, and monitor for safety and efficacy subjects who have previously received a BCMA-targeted therapy as a separate line of therapy potentially in a separate clinical trial. Additionally, several |

| Protocol Revision Chronology: | |
|---|---|
| | eligibility criteria were updated, clarification was made that enrolment into Arm 2 only (versus both arms) would be paused following start of lymphodepletion of the third subject, and the version of International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma used in efficacy determination was updated from 2011 to 2016. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Change to Protocol Specified Statistical Analysis Plan

In this RAP, there are no changes or deviations to the statistical analysis from that described in the latest amended protocol (dated 24-Feb-2020) other than the following:

- Definitions of analysis populations, removing the As-Treated Population.
- Explicit instruction to summarize data for the Modified Intent-to-Treat (mITT) Population (instead of Intent-to-Treat [ITT] Population), when the two populations are identical.
- Efficacy endpoints described in the Efficacy Analyses section (Section 7) as Primary and Secondary Efficacy Endpoints, rather than overall Secondary Endpoints.
- Protocol Section 11.2 states that "Interim analyses to inform internal decision making may be performed for each arm after enrolment to the arm is complete and all enrolled subjects in that arm who will receive NY-ESO-1<sup>c259</sup>T have done so and of those: all have completed at least three disease assessments since infusion or have progressed (And if progressed prior to the Week 9 visit have been followed up for safety for a minimum of 9 weeks following T-cell infusion) or have died or were withdrawn from the study." As accrual to the study was halted prior to completing enrolment in either arm, the interim analysis was not conducted. Thus, references to the interim analysis and the evaluable population have been removed from the RAP.
- Protocol Section 3.1.3 and Section 4.3 state that "A subject will be considered to have completed the treatment phase of the study when he/she has progression of disease or 108 weeks after NYESO-1<sup>c259</sup>T-cell infusion, whichever is sooner". In this RAP, death is also considered a criterion for completion of the treatment phase.
- Protocol Section 4.4 states that "This study will be considered complete when the last subject has been rolled over into the LTFU protocol." This RAP notes that study completion can also occur in the case that one or more patients have withdrawn from the parent study (including lost to follow-up), completed long-term follow-up in this study, or expired prior to rolling over into the LTFU protocol.
- Protocol Section 6.1 states that "Subjects receiving any of palliative radiation therapy that could be foreseen impacting disease course or disease assessments will be censored for the purposes of determining PFS." In this RAP, new anti-cancer therapy that would result in censoring PFS only includes systemic therapy.
- This study was terminated early; thus, only analyses relevant to these limited data are presented.
- Due to early termination of the study, only a final analysis will be performed. Thus, a primary analysis has been removed from Section 3.
- According to GSK standards, Listing of Race (DM9) is required per ICH E3. Due to differences in Adaptimmune data collection, only Listing of Demographic Characteristics (DM2) will be displayed which will include race information.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| • To describe the safety and tolerability of autologous genetically modified T-cells (NY-ESO-1c259T) alone (Arm 1) or in combination with pembrolizumab (Arm 2) in participants who are human leukocyte antigen HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 positive and have NY-ESO-1 and/or LAGE-1a positive relapsed refractory multiple myeloma (RRMM). | Adverse events (AEs and Treatment<br>Limiting Toxicity (TLT) rate),<br>including serious adverse events<br>(SAEs); laboratory assessments,<br>including chemistry, hematology,<br>and coagulation; and cardiac<br>assessments by electrocardiogram<br>(ECG). |
| Secondary Objectives | Secondary Endpoints |
| To describe the antitumor activity of autologous genetically modified T-cells (NY-ESO-1c259T) alone (Arm 1) or in combination with pembrolizumab (Arm 2) in participants who are HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 positive and have NY-ESO-1 and/or LAGE-1a positive RRMM. | <ul> <li>Overall Response Rate (ORR).</li> <li>Time to Response (TTR).</li> <li>Duration of Response (DoR) for participants who achieve at least a Partial Response (PR).</li> <li>Progression-free survival (PFS).</li> </ul> |
| To describe persistence of autologous genetically modified T-cells (NY-ESO-1c259T) over time. | Maximum persistence (Cmax), time to Cmax (Tmax), and area under the time curve from zero to time t (AUC(0-t)), as data permit. |

| <b>Exploratory Objectives</b> | <b>Exploratory Endpoints</b> |
|---|---|
| • To describe the antitumor activity of autologous genetically modified T-cells (NY-ESO-1 <sup>c259</sup> T) alone (Arm 1) or in combination with pembrolizumab (Arm 2) in participants who are HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 positive and have NY-ESO-1 and/or LAGE-1a positive RRMM. | Overall survival (OS). |
| To evaluate minimal residual disease<br>(MRD) at 4 months post T-cell infusion<br>(Week 15). | MRD Rate at Week 15. |
| • To evaluate the persistence, phenotype, and functionality of NY-ESO-1 <sup>c259</sup> positive T-cells. | • Correlate persistence, phenotype, and functionality of NY-ESO-1 <sup>c259</sup> T in the peripheral blood and/or bone marrow with response to treatment and safety. |
| To understand mechanisms of resistance to NY-ESO-1 <sup>c259</sup> T. | <ul> <li>Determine whether loss of NY-ESO-1 and/or LAGE-1a expression in myeloma cells is a resistance mechanism.</li> <li>Correlate apparition of anti-NY-ESO-1<sup>c259</sup>T antibodies with efficacy and safety.</li> <li>Correlate expression of PD-L1 in the tumor microenvironment and PD-1 expression on T-cells with response to treatment.</li> <li>Correlate frequency of immune cell subsets in peripheral blood and/or bone marrow with treatment response.</li> <li>Correlate frequency of immune cell subsets in peripheral blood and in bone marrow.</li> </ul> |
| To evaluate antigen spreading as a mechanism of response. | Correlate clonal outgrowth of T-cell populations with tumor response following T-cell infusion. |
| To evaluate cytokine levels pre- and post-infusion on cytokine release syndrome (CRS). | Correlate cytokine levels with incidence and severity of CRS or other safety events. |
| • To evaluate the impact of germline polymorphisms in IL-6, TNF-α, IL-10, IFN-γ and TGF-β on CRS. | Correlate polymorphisms in germline deoxyribonucleic acid (DNA) with CRS. |

# 208470

# 2.3. Study Design

# **Overview of Study Design and Key Features**



#### **Overview of Study Design and Key Features**

## Design Features

- This is a 2-arm, open-label, pilot study, with 3 distinct parts: (1) Eligibility Screening, (2) Leukapheresis/Manufacturing, and (3) Lymphodepletion/Treatment, with Parts 2 and 3 collectively representing the Treatment Phase.
- Participants will first undergo screening for HLA-type (HLA-A\*02:01, HLA-A\*02:05, and/or HLA-A\*02:06) and presence of antigen NY-ESO-1 and/or LAGE-1a in their bone marrow. Only participants who are selected after HLA-genotyping and determination of antigen expression will be considered for further eligibility screening.
- In the initial study design, participants meeting all eligibility criteria were assigned to 1 of 2 treatment arms: NY-ESO-1<sup>c259</sup>T alone (Arm 1) or NY-ESO-1<sup>c259</sup>T in combination with pembrolizumab (Arm 2). Following protocol amendment 5, the enrolment of participants in Arm 1 will be completed before the enrolment of participants in Arm 2 continues.
- Following enrolment, participants will undergo leukapheresis to obtain cells for the manufacture of autologous NY-ESO-1<sup>c259</sup> bearing T-cells.
- When NY-ESO-1<sup>c259</sup>T-cells are available, participants will undergo lymphodepleting chemotherapy with fludarabine and cyclophosphamide and receive granulocyte-colony stimulating factor (G-CSF) support before undergoing infusion of NY-ESO-1<sup>c259</sup>T-cells.
- Re-confirmation of eligibility and baseline assessments will occur during the 7 days preceding lymphodepleting chemotherapy.
- Participants may receive anticancer therapy between screening and leukapheresis and between leukapheresis and lymphodepletion, with mandatory wash-out periods respected.
- Ten participants per arm (20 participants in total) are targeted to be enrolled in the study and receive the NY-ESO-1<sup>c259</sup>T infusion, with at least 6 participants per arm having received and failed BCMA-based therapy (CAR-T, ADC, or other types of BCMA-targeted therapies) between screening and leukapheresis and/or between leukapheresis and lymphodepletion.
- Eligible participants who do not receive the NY-ESO-1<sup>c259</sup>T infusion for any reason will be replaced, and infused participants in Arm 2 who do not receive pembrolizumab will be included in Arm 1 for purposes of analysis and replaced within Arm 2. Analyses describing the Intent-to-Treat (ITT) population will summarize by the treatment group to which the participant was assigned.
- A participant will be considered to have completed the treatment part of the study at the earliest of confirmed disease progression (with minimum 9 weeks of follow-up for safety), 108 weeks after NY-ESO-1<sup>c259</sup>T-cell infusion, or death.

| Overview of Str | udy Design and Key Features |
|---|---|
| | • After treatment, participants will be rolled into a long-term follow-up (LTFU) study under a separate protocol and followed at month 3, 6, and 12, then every 6 months for 5 years, and then yearly for up to 15 years. If the LTFU protocol is not available, follow-up will start on this protocol following the guidelines listing above until the LTFU becomes available. |
| Dosing | <ul> <li>The 2 investigational products (IPs) in this study are: <ul> <li>NY-ESO-1<sup>c259</sup>T: An autologous T-cell transduced with a self-inactivating lentivirus encoding for a high affinity NY-ESO-1/LAGE-1a-specific T-cell receptor (TCR), administered through a single IV infusion (cell range: 1 × 10<sup>9</sup> to 8 × 10<sup>9</sup> transduced cells) in both treatment arms.</li> <li>Pembrolizumab: A humanized monoclonal antibody, administered as a fixed dose of 200 mg through a 30-minute IV infusion in Arm 2.</li> </ul> </li> <li>Participants in both arms who have been re-confirmed as eligible during the baseline assessment period (Day -14 to -8) will undergo lymphodepleting chemotherapy with fludarabine (30 mg/m²/day) on Days -8, -7, -6, and -5 and cyclophosphamide (900 mg/m²/day) on Days -7, -6, and -5, followed by G-CSF support on Day -4 and infusion of NY-ESO-1<sup>c259</sup>T-cells on Day 1.</li> <li>For participants in Arm 2, pembrolizumab will be administered on Day 22 (Week 3; 21 days after NY-ESO-1<sup>c259</sup>T infusion) and then every 3 weeks thereafter up to Week 108. If the participant experiences toxicity preventing Week-3 dosing of pembrolizumab, the first dose of pembrolizumab may be administered on Week 6 instead. If toxicity still prevents starting pembrolizumab dosing at Week 6, the participant will not be administered pembrolizumab and</li> </ul> |
| Time & | <ul> <li>will be followed as a participant in Arm 1.</li> <li>Refer to Appendix 2: Schedule of Activities</li> </ul> |
| Events | |
| Treatment<br>Assignment | Participants meeting all eligibility criteria will be treated in one of two treatment arms: |
| | <ul> <li>Arm 1: Participants will receive NY-ESO-1<sup>c259</sup>T alone as a single infusion on Day 1, 4 days after completing fludarabine, cyclophosphamide, and G-CSF (there is no Day 0 for this study).</li> <li>Arm 2: Participants will receive NY-ESO-1<sup>c259</sup>T in combination with pembrolizumab. NY-ESO-1<sup>c259</sup>T will be administered as a single infusion on Day 1, 4 days after completing fludarabine, cyclophosphamide, and G-CSF. Pembrolizumab will be administered first on Day 22 (Week 3) and then every 3 weeks thereafter up to Week 108.</li> <li>Eligible participants who do not receive the NY-ESO-1<sup>c259</sup>T infusion for any reason will be replaced, and infused participants in Arm 2 who do not receive pembrolizumab will be included in Arm 1 for</li> </ul> |

| Overview of Stu | udy Design and Key Features |
|---|---|
| | <ul> <li>purposes of analysis and replaced within Arm 2. Analyses describing the Intent-to-Treat (ITT) population will summarize by the treatment group to which the participant was assigned.</li> <li>The study initially was initially designed to randomize participants to the two arms. Following protocol amendment 5, the enrolment of participants in Arm 1 will be completed before the enrolment of participants in Arm 2 continues.</li> </ul> |
| Safety | Safety will be assessed at each clinic visit. A Safety Review Team |
| Monitoring | (SRT) may review safety data in both treatment arms at any time. |
| Review for | TLTs will be evaluated for participants in Arm 2 only. |
| TLTs | • Enrolment in Arm 2 will be paused after the third enrolled |
| | <ul> <li>participant has initiated lymphodepleting chemotherapy. A complete safety review of the first 3 Arm 2 participants will be conducted before enrolment resumes.</li> <li>The SRT may recommend pausing the study at any time to evaluate safety and, if warranted, to close an arm of the trial (e.g., in Arm 2, if at an interim assessment the predictive probability that the TLT rate for participants exceeds 33%, is greater than 50%).</li> <li>Interim analyses to inform internal decision-making may be performed for each arm after enrolment to the arm is complete and all enrolled participants in that arm who will receive NY-ESO-1<sup>c259</sup>T have done so and have completed at least 3 disease assessments since infusion, progressed (if progressed prior to Week 9, then have been followed for safety for at least 9 weeks following infusion), died, or withdrawn from the study. Additional analyses may be undertaken when all participants in Arm 1 satisfy the criteria for primary analysis. Given accrual to the study was stopped prior to completing enrolment to either arm, this interim analysis will not occur.</li> </ul> |

# 2.4. Statistical Analyses

This study is not powered to compare safety or efficacy between the 2 treatment arms. Therefore, no hypothesis testing or formal statistical comparisons are planned. All analyses will be descriptive in nature. Continuous data will be summarized, minimally, using n, means, medians, standard deviations, and ranges, while categorical data will be summarized using frequency counts and percentages or proportions. Graphical summaries of the data will be presented, as appropriate. Time-to-event endpoints will be summarized as the median and 25th and 75th percentiles and displayed graphically using Kaplan-Meier (product-limit) curves, if the data warrant.

## 3. PLANNED ANALYSES

# 3.1. Safety Monitoring Review for TLTs

After the third participant in Arm 2 has initiated lymphodepleting chemotherapy, enrolment will be paused. Enrolment may resume after these participants have received both T-cells and pembrolizumab and a complete safety review by the SRT of Treatment-Limiting Toxicities (TLT) has been conducted.

Additionally, safety review for the assessment of TLTs may be carried out at any time in Arm 2. The SRT may recommend pausing the study to evaluate safety and, if warranted, stopping the trial (e.g., if the predictive probability of the TLT rate exceeding 33% is greater than 50%).

#### 3.1.1. Predictive Probabilities

Predictive probabilities will be estimated for participants in Arm 2 only.

As participants are accrued and at  $n\ge3$  participants, Bayesian predictive probabilities will be used to evaluate TLTs in Arm 2. If, the probability of the end-of-trial TLT rate exceeding 0.33 is greater than 0.50 at an interim assessment (i.e., when n < [Nmax = 10]), then the SRT may recommend to pause the study for safety review and, if warranted, to stop the trial for safety.

To evaluate the TLT rate using a Bayesian framework, let p denote the TLT rate for Arm 2, and let X denote the number of TLTs in  $n\ge3$  participants. X is assumed to follow a binomial distribution B(n, p). Assuming a non-informative prior distribution of beta (0.18, 0.82) for the TLT rate, the posterior of the TLT rate will follow a beta (0.18+x, 0.82+n-x) distribution.

Let Y represent the number of TLTs in m (equal to  $N_{max} - n$ ) future participants. With the aforementioned prior and likelihood, Y follows a beta-binomial (m, 0.18+x, 0.82+n-x) distribution. This distribution will be explored to better estimate the probability of observing y (0 [zero] to m) TLTs in the m future participants.

Let the predictive probability (PP) equal the probability of the end-of-trial TLT rate exceeding 0.33, given the maximum planned sample size (N<sub>max</sub>) of 10. Using results from the first n participants, a defined  $\theta$ =0.9, and methods described by Lee and Liu (Lee, 2008), PP will be computed as the weighted average (i.e., weighted by the probability of the realization of each Y) as? the indicator of a positive trial (i.e., at each Y, the probability of TLT rate > 0.33 is greater than 90%), should the current trend continue and the trial be conducted until the end of the study.

Refer to Table 1 below for the calculated PP associated with  $n < N_{max}$ . If at least 2 of the first 3 participants experience a TLT, the trial should be paused to further evaluate safety. Similarly, the trial may be paused for safety evaluation if at least 3 of the first 4 or 5 participants, at least 4 of the first 6 or 7 participants, or at least 5 of the first 8 or 9 participants experience a TLT.

Table 1 Predictive Probabilities for  $N_{max} = 10$ 

| | X=0 | X=1 | X=2 | X=3 | X=4 | X=5 | X=6 | X=7 | X=8 | X=9 |
|---|---|---|---|---|---|---|---|---|---|---|
| n=3 | 0.0017 | 0.115 | 0.566 | 0.9426 | NA | NA | NA | NA | NA | NA |
| n=4 | 0.0002 | 0.0341 | 0.3083 | 0.7812 | 0.9842 | NA | NA | NA | NA | NA |
| n=5 | 0 | 0.0059 | 0.1255 | 0.5447 | 0.9165 | 0.9974 | NA | NA | NA | NA |
| n=6 | 0 | 0 | 0.0298 | 0.2932 | 0.7678 | 0.9813 | 1 | NA | NA | NA |
| n=7 | 0 | 0 | 0 | 0.0956 | 0.5305 | 0.9279 | 1 | 1 | NA | NA |
| n=8 | 0 | 0 | 0 | 0 | 0.2406 | 0.7954 | 1 | 1 | 1 | NA |
| n=9 | 0 | 0 | 0 | 0 | 0 | 0.518 | 1 | 1 | 1 | 1 |

Furthermore, if the threshold exceeds 0.5, as described above, other supportive information may be computed. For example, the PP distribution may also be evaluated to calculate the probabilities associated with specific outcomes. For instance, if 4 of 7 participants experience a TLT, then the beta-binomial (3, 4.18, 3.82) will be used to compute the probability of observing TLTs in 1 or more of the remaining 3 participants, the average number participants with at least one TLT, the variability around these estimates, etc. In addition, the 95% credible interval for the TLT rate will be derived from the posterior distribution. These and other characteristics of the posterior distribution and posterior predictive distribution may aid in the evaluation of TLT rates.

# 3.2. Interim Analyses

Protocol Section 11.2 states that interim analyses to inform internal decision-making may be performed for each arm after enrolment to the arm is complete and all enrolled participants in that arm who will receive NY-ESO-1<sup>c259</sup>T have done so and have completed at least 3 disease assessments since infusion, progressed (if progressed prior to Week 9, then have been followed for safety for at least 9 weeks following infusion), died, or withdrawn from the study. Additional analyses may be undertaken when all participants in Arm 1 satisfy the criteria for primary analysis.

Note that such an interim analysis is not planned and thus is not listed as a deliverable in Appendix 12: List of Data Displays.

208470

# 3.3. Final Analysis

The final analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study or have withdrawn from the study for any reason. A participant will complete the treatment phase of the study upon disease progression, death, or 108 weeks after NY-ESO-1<sup>c259</sup>T-cell infusion, whichever is sooner. All infused participants will enter a LTFU protocol. Study completion occurs when all participants in the treatment phase of the study have rolled over to the LTFU protocol GSK208750 (ADP-0000-002), completed long-term follow-up in this study, expired, or withdrawn (including lost to follow-up) from the parent study before rollover to the LTFU protocol
- 2. All required database cleaning activities have been completed and final DBR and DBF has been declared by Data Management.

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who signed the screening informed consent form. | Screen failures |
| Enrolled | All participants who underwent<br>leukapheresis, with treatment arm<br>identified as the assigned<br>(planned) arm. | <ul> <li>Required study<br/>population displays<br/>(see Appendix 12:<br/>List of Data Displays<br/>for specific displays)</li> </ul> |
| Intent-To-<br>Treat (ITT) | • All participants who underwent leukapheresis, with treatment arm identified as the assigned (planned) arm. | <ul><li>Study population</li><li>Primary safety (where appropriate)</li></ul> |
| Modified<br>Intent-To-<br>Treat (mITT) | • All participants in the ITT Population who received the NY-ESO-1 <sup>c259</sup> T infusion, with treatment arm identified as the arm of actual treatment received. | <ul><li>Efficacy</li><li>Primary safety (where appropriate)</li></ul> |

Refer to Appendix 12: List of Data Displays, which details the population to be used for each display. Note that, if an analysis is planned for both the mITT and ITT Population and these populations contain the same participants in the same arms, then results will be reported for the mITT Population only.

#### 4.1. Protocol Deviations

Protocol deviations will be tracked in accordance with the Protocol Deviation Specification Form by the study team throughout the conduct of the study and sent to the Data Manger and Biostatistics Lead in a spreadsheet. Protocol deviations will not be identified programmatically.

Inclusion/exclusion criteria deviations will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Data will be listed and summarized according to GSK reporting standards, as applicable.

# 5.1. Study Treatment & Sub-group Display Descriptors

Two treatment arms are included in this study (Arm 1: Participants who receive NY-ESO-1<sup>c259</sup>T alone; Arm 2: Participants who receive NY-ESO-1<sup>c259</sup>T in combination with pembrolizumab). As data will be displayed within summaries and listings principally by treatment arm, the table below provides an example of the treatment descriptors to be used for distinguishing the treatment arms within the displays. Actual treatment doses may differ (e.g., in the case of modified pembrolizumab dosage) but will follow the same format.

| Treatment Group Descriptions | |
|------------------------------|---|
| Data Displays for Reporting | |
| Description Order in TLF | |
| GSK794 | 1 |
| GSK794+PEMBRO | 2 |
| Total 3 | |

All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

## 5.2. Baseline Definitions

Unless otherwise specified, baseline values will be represented by the latest non-missing measurements (including unscheduled visits) prior to the start of lymphodepleting chemotherapy. Per protocol, baseline assessments should occur within the 7 days preceding lymphodepletion. If an assessment is not performed within the 7-day window, then the latest assessment prior to the 7-day window will be used. If an assessment is performed on the same date as the start of lymphodepletion and the time of assessment is not recorded, then the assessment will be assumed to have occurred prior to lymphodepletion and used as baseline.

For ECG parameters, if baseline values are missing (given the aforementioned baseline definition of latest record within the 7 days preceding lymphodepletion), then baseline values will be represented by the mean of values recorded during the screening and Day 1 pre-dose assessments.

For participants who do not receive lymphodepleting chemotherapy during the study, baseline values will be represented by the latest, non-missing measurements recorded. If baseline data is missing, then no derivation will be performed, and baseline will be set to missing.

## 5.3. Multicentre Studies

Data from all participating centres will be pooled prior to analyses.

It is anticipated that participant accrual will be spread thinly across centres. Consequently, data summaries by centre are unlikely to be informative and will not be provided.

# 5.4. Examination of Covariates, Other Strata and Subgroups

No covariates or strata will be incorporated into analyses, and no subgroup analyses will be performed in this study.

# 5.5. Multiple Comparisons and Multiplicity

No formal statistical testing will be performed; therefore, no adjustments for multiple comparisons or multiplicity are planned.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the following appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 14.3 | Appendix 3: Assessment Windows |
| 14.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 14.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 14.6 | Appendix 6: Derived and Transformed Data |
| 14.7 | Appendix 7: Reporting Standards for Missing Data |
| 14.8 | Appendix 8: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

Study population analyses will be based on the ITT Population, unless otherwise specified. Some study population analyses will be repeated in the mITT population. If the mITT and ITT Populations contain the same participants in the same arms, then results planned for both the ITT & mITT populations will only be reported for the mITT Population.

Based on GSK Core and Oncology Data Standards, study population analyses will include summaries and listings of participant disposition, protocol deviations, demographic and other baseline characteristics, prior and concomitant medications, study treatment exposure, disease characteristics at initial diagnosis and screening, and prior and on-study anti-cancer therapies, prior anti-cancer radiotherapy, and prior and on-study surgical procedures. Details of the planned displays are presented in Appendix 12: List of Data Displays.

# 6.2. Disposition of Participants

Using the Screened Population, a summary and a listing of screening status and reasons for screen failure will be provided. A summary of the number of participants in each analysis population (see Section 4 for definitions) and a listing of participants excluded from each population will also be provided detailing reason for exclusion.

Overall study disposition, including transfer to the separate LTFU protocol GSK208750, will be summarized.

Treatment phase status for both arms will be summarized with reasons for non-completion as captured in the eCRF.

Listings of data describing reasons for study withdrawal and study treatment status will be produced, with the latter including dates and times, associated with leukapheresis, lymphodepletion, and T-cell infusion, dose level of T-cell infusion, indicators of treatment phase completion (vs. discontinuation), end of study status, and reasons for treatment phase discontinuation.

A summary and listing of pembrolizumab treatment status and reasons for discontinuation will be generated for participants in Arm 2.

Lastly, the number of participants in the Enrolled Population will be listed by country and study site ID.

#### 6.3. Protocol Deviations

Important protocol deviations will be summarized and listed.

A separate listing of inclusion/exclusion deviations will also be provided.

# 6.4. Demographic and Baseline Characteristics

Demographic characteristics, including race, age, ethnicity, sex, height, baseline body weight, body mass index (BMI), and body surface area (BSA) as per the Mosteller formula, will be both summarized and listed. Age, height, weight, BMI, and BSA will be summarized as continuous variables, while age, sex, race, and ethnicity will be summarized as categorical variables. Age will be categorized and summarized using the GSK IDSL standard (≤18, 19-64, and ≥65 years), and in a separate summary, using EudraCT (18-64, 65-84 and ≥85 years). Age will be derived per Section 14.6.2.

Separate summaries and listings of disease characteristics at initial diagnosis and at screening will be provided. Disease characteristics including time from initial diagnosis to screening ICF signed (in months), stage at diagnosis, histologic type, percent clonal bone marrow plasma cells, presence and type of end organ damage, presence and type of plasmacytoma, presence of bone lesion(s), and chromosomal aberrations will be summarized and listed. Disease characteristics at screening will include type of multiple myeloma, HLA-A status, NY-ESO-1 status, LAGE-1a status, number of systemic therapy regimens prior to leukapheresis, number of radiotherapy regimens prior to leukapheresis, receipt of stem-cell transplant prior to leukapheresis (Y/N), and subtype of stem-cell transplant received (autologous or allogeneic). Listings will additionally disclose relevant dates (e.g., diagnosis date, dates of antigen testing). Derivation of the number of prior systemic therapy regimens should include therapies recorded as systemic therapy, as well as stem cell therapy and associated conditioning chemotherapy as a prior line. Time from initial diagnosis to screening ICF signed (in months) will be calculated as detailed in Appendix 6.

Medical conditions (history and ongoing) at screening will be listed and summarized.

#### 6.5. Prior and Concomitant Medications

All concomitant medications will be summarized (for the mITT Population only), and all prior and concomitant medications will be included in a single listing. The definitions of prior and concomitant medications are provided in Appendix 4: Study Phases and Treatment Emergent Events.

Medications will be coded using GSK Drug coding dictionary. The summary of concomitant medications will show the number and percentage of participants taking concomitant medication by Ingredient. Multi-ingredient products will be summarized by their separate ingredients rather than as a combination of ingredients. Anatomical Therapeutic Chemical (ATC) classification Level 1 (Body System) information will be included in the dataset created but will not appear on the listing or summary.

In the summary of concomitant medications, each participant will be counted once per unique ingredient. For example, if a participant takes Amoxycillin on 2 separate occasions, the participant will be counted only once under the ingredient "Amoxycillin". In the summary of concomitant medications, ingredients will be summarized by the base only.

Data describing concomitant receipt of blood products will be both summarized and provided in a listing.

# 6.6. Study Treatment Exposure

Study treatments – described in Section 5 of the protocol – are leukapheresis, lymphodepleting chemotherapy, NY-ESO-1<sup>c259</sup>T cell infusion, and pembrolizumab.

The number and percentage of participants having undergone leukapheresis, lymphodepleting chemotherapy, T-cell infusion (overall and given the minimum dose of  $1 \times 10^9$  transduced cells), and pembrolizumab infusion will be summarized.

The total number of transduced T-cells will be summarized as both a continuous variable and categorical variable. Categories will include <1, 1 to  $\le$ 8, and >8 (x 10<sup>9</sup> cells) and <1, 1 to  $\le$ 3, >3 to  $\le$ 8, and >8 (x 10<sup>9</sup> cells). An associated listing will provide T-cell infusion start/stop dates/times (over all bags), average vector copy number per cell in cell product, total number of transduced cells, and percentage of cells transduced.

For participants in Arm 2, pembrolizumab dose intensity (mg/3 weeks) and number of pembrolizumab cycles received will be listed. A listing, disclosing the details of pembrolizumab exposure, will also be generated. Additionally, a listing will be provided for all dose delays experienced on the study and duration of delay. Duration of delays is defined as period from the expected start date of dose to actual start date of current dose. The calculation of duration of delay is actual start date of current dose - expected start date of dose. Expected start date of dose = actual start date of previous dose + 21. Note that the expected start date of the first dose of pembrolizumab is 21 days after T-cell infusion. Thus, if this dose is not received, this will be considered a dose delay.

Dose administration data for lymphodepleting chemotherapy, including fludarabine and cyclophosphamide, will be presented in a single data listing. Lastly, a single participant-level data listing will be dedicated to disclosing dates of leukapheresis, lymphodepleting chemotherapy, T-cell infusion, and pembrolizumab infusion.

# 6.7. Anti-Cancer Therapies

Number and percentage of participants who receive any anti-cancer therapy (including systemic therapy and radiotherapy) or cancer-specific surgery will be provided in separate summaries. Systemic therapy drugs will be coded using the GSK Drug coding dictionary, then summarized by ingredient. Participant-level data describing all anti-cancer therapies and cancer-specific surgeries will be provided in separate listings.

#### 6.7.1. Prior Anti-Cancer Therapies

Anti-cancer therapies will be classified into prior and on-study phases as described in Appendix 4. Note that only therapies initiated on or after the first day of lymphodepletion chemotherapy are considered on-study. Prior therapies will be further classified into subphases at date of leukapheresis.

Prior therapy types will include systemic therapy (including stem cell therapy), radiotherapy, and cancer-related surgery, with systemic therapies other than stem cell therapy coded using the GSK Drug coding dictionary. While all therapy types will be described within each of the aforementioned summaries, the details of each therapy type will be provided in separate listings.

Summaries of the numbers of radiotherapy and systemic anti-cancer regimens received prior to leukapheresis will be presented as part of the summary of disease characteristics at screening.

Systemic anti-cancer therapy regimens initiated between leukapheresis and lymphodepletion (as defined in Appendix 4) will be categorized as either bridging (regimens administered to maintain/stabilize the participant until T-cell infusion) or full lines (regimens administered with the intent of disease effect) by GSK physician review.

Bridging therapies will be excluded from summaries of prior anti-cancer therapy.

Thus, unless otherwise stated, summaries of prior systemic anti-cancer therapies will include all therapies before lymphodepletion except those in the leukapheresis to lymphodepletion period identified as bridging therapies. (Note that this is equivalent to all therapies prior to leukapheresis plus therapies initiated between leukapheresis and lymphodepletion identified as full lines.)

A breakdown of the number of participants who received each type of prior anti-cancer therapy will be presented.

Anti-cancer therapy will be coded using GSK Drug coding dictionary. The number of participants receiving prior anti-cancer therapies will be summarized by ATC Level 1 and ingredient. Bridging therapies will be similarly summarized.

A summary of the number of overall systemic prior anti-cancer therapy regimens and radiotherapies prior to lymphodepletion will also be produced. Systemic therapy regimens will not be broken down by type of systemic therapy since different types of therapies are expected within a regimen.

All prior anti-cancer therapy will be listed with subphase indicated and bridging therapies flagged.

All anti-cancer radiotherapy (including on-study) will be listed, with phase and subphase indicated.

All prior cancer related surgical procedures will be listed, with subphase indicated. Those before lymphodepletion will be summarized by intent and site.

## 6.7.2. On-Study Anti-Cancer Therapies

The number and percentage of participants who receive any anti-cancer therapy (including systemic therapy, radiotherapy, and stem cell therapy) or cancer-specific surgery will be provided in separate summaries. Systemic therapy drugs will be coded

208470

using the GSK Drug coding dictionary, then summarized by ingredient. Participant-level data describing all anti-cancer therapies and cancer-specific surgeries will be provided in separate listings.

#### 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Analyses

All efficacy analyses are planned to be performed by treatment arm and overall. Efficacy Analyses will be conducted according to International Myeloma Working Group (IMWG) (2016) Criteria [Kumar 2016, Section 13].

## 7.1.1. Primary Endpoint/Variable: Overall Response Rate (ORR)

With minimal exception (see description of Confirmed Response below), only disease assessments occurring from the start of NY-ESO-1<sup>c259</sup>T infusion to the earlier of confirmed progressive disease (PD) or initiation of new anti-cancer therapy (including only systemic therapy) will be considered. Note that while considered a primary endpoint for the purposes of efficacy analysis in this RAP, ORR is defined as a secondary objective in the protocol.

#### 7.1.1.1. Best Overall Response

The BOR is defined as the best confirmed response (stringent Complete Response [sCR] > Complete Response [CR] > Very Good Partial Response [VGPR] > Partial Response [PR] > Minimal Response [MR] > Stable Disease [SD] > Progressive Disease [PD] > Not Evaluable [NE]) from treatment start date until disease progression or initiation of new anti-cancer therapy (including only systemic therapy), whichever is earlier, as assessed per IMWG (2016). Participants with only assessments of not evaluable (NE) or missing response will be treated as non-responders (i.e., they will be included in the denominator when calculating BOR percentages and the proportion representing ORR).

#### 7.1.1.2. Overall Response Rate

The primary efficacy endpoint is ORR, defined as the percentage of participants with a best overall response (BOR) of confirmed stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) per IMWG (2016). Details regarding derivation of confirmed response are provided in Table 2.

#### 7.1.1.3. Definition of Adequate Assessment

An adequate assessment for purposes of identifying BOR and computing ORR is defined as a disease assessment with Investigator-assessed response of sCR, CR, VGPR, PR, MR, SD, or PD per IMWG (2016). This definition of adequate assessment differs from that used for time-to-event endpoints (see Section 7.2, Secondary Efficacy Analyses).

#### 7.1.1.4. Date Associated with Response

A disease assessment may occur at a scheduled or unscheduled visit. While the date of assessment recorded on the Disease Assessment eCRF may or may not exactly match the dates of all procedures supporting the assessment and associated with the visit, it will be used to represent the date of response.

#### 7.1.1.5. Confirmed Response

An individual Investigator-assessed response must be confirmed at a subsequent disease assessment. Details describing the derivation of a confirmed response are provided below and in Table 2.

Pertaining to the responses of sCR, CR, VGPR, PR, and MR, a confirmed response is an Investigator-assessed response that has been documented at the confirmed response level or better across 2 consecutive adequate disease assessments (referred to as "first assessment" and "subsequent assessment"). First and subsequent disease assessments are consecutive, representing a dual-assessment scenario. The subsequent assessment is defined as the next adequate assessment (i.e., not missing or with NE response) following the first assessment, before (or on the same date of) start of new anti-cancer therapy (except for confirmation of PD, for which PD or death due to disease under study after new anti-cancer therapy may be confirmation of PD). No minimal time interval is required for the subsequent disease assessment, but a different sample is required for confirmation. If 2 consecutive assessments are performed on different dates, the assumption will be made that the 2 assessments are based on different samples.

• Note that, for participants who receive subsequent anti-cancer therapy, no imputation will be performed for completely missing start dates. However, if the start date of the anti-cancer therapy is partial (i.e., either missing the day but has the month and year available or missing both day and month), then the imputation rules described in Section 14.7.2.1, Handling of Missing and Partial Dates, will be applied.

 Table 2
 Response Confirmation Algorithm

| Response Documented at<br>the First Assessment <sup>[1]</sup> | Response Documented at the Subsequent Assessment | Confirmed Response Associated with the First Assessment <sup>[1]</sup> |
|---|---|---|
| sCR | sCR | sCR |
| sCR | CR | CR |
| CR | sCR/CR | |
| sCR/CR | VGPR | VGPR |
| VGPR | sCR/CR/VGPR | |
| sCR/CR/VGPR | PR | PR |
| PR | sCR/CR/VGPR/PR | |
| sCR/CR/VGPR/PR | MR | MR |
| MR | sCR/CR/VGPR/PR/MR | |
| sCR/CR/VGPR/PR/MR/SD | SD/PD/NE | |
| | <u>OR</u> | |
| | No subsequent disease assessment prior | SD |
| | to new anti-cancer therapy, if any | SD |
| | (participant may or may not still be on | |
| | study) | |
| PD (due to reasons other | PD (any reason), including PD after | PD |
| than imaging, i.e., | initiation of new anti-cancer therapy | |
| plasmacytoma or bone | <u>OR</u> | |
| lesion) | | |

| Response Documented at the First Assessment <sup>[1]</sup> | Response Documented at the Subsequent Assessment | Confirmed Response Associated with the First Assessment <sup>[1]</sup> |
|---|---|---|
| | No subsequent disease assessment: participant died due to disease under study before further adequate assessment could be performed (including death due to disease under study after initiation of new anti-cancer therapy) | |
| PD due to imaging (i.e., plasmacytoma or bone lesion) | Any OR No subsequent disease assessment | |
| PD (due to reasons other than imaging, i.e., plasmacytoma or bone lesion) | sCR/CR/VGPR/PR/MR/SD OR No subsequent disease assessment | NE |
| NE or missing | Any OR No subsequent disease assessment | |

<sup>&</sup>lt;sup>1</sup> The date of confirmed response for all scenarios equals the date associated with the first disease assessment.

# 7.1.2. Summary Measurement

The number and percentage of participants in the following best confirmed response categories will be summarized: sCR, CR, VGPR, PR, overall response (sCR+CR+VGPR+PR), MR, SD, PD, and NE. Corresponding 2-sided exact (Clopper-Pearson) 95% CIs for ORR will also be provided for each arm and total. Participants with unknown or missing responses will be considered NE.

A participant-level data listing of Investigator-assessed responses per assessment timepoint, visit level response, and BOR will be provided, including the name of the corresponding visit, date of the response assessment, study day, and observed response.

A spider plot for the change from baseline over time and a waterfall plot showing the maximum percent reduction from baseline will be produced for Serum M-protein, Urine M-protein and Serum free light chain (FLC), if data warrant. The maximum percent reduction will be plotted in the following hierarchical order:

- (1) Plot Serum M-protein maximum percent reduction from baseline, if data are available:
- (2) If (1) is not feasible, plot Urine M-protein maximum percent reduction from baseline, if data are available;
- (3) If both (1) and (2) are not feasible, plot maximum percent reduction from baseline for difference between 2 types of Serum FLC, if data are available.

#### Difference between 2 types of Serum FLC

The percent change from baseline for difference between 2 types of Serum FLC is defined as:

(post-baseline difference – baseline difference) / baseline difference x 100.

To calculate the difference, the "involved" and "non-involved" light chains must be determined first, based on the ratio of non-missing values for Serum Kappa FLC protein and Serum Lambda FLC protein at baseline.

The detailed algorithm is provided as below:

- If the baseline ratio of (Kappa FLC/Lambda FLC) > 1.65, then Kappa FLC is defined as involved FLC, and Lambda FLC is defined as non-involved FLC. Then:
  - o Difference between involved and uninvolved = Kappa FLC Lambda FLC.
- If the baseline ratio of (Kappa FLC/Lambda FLC) < 0.26, then Lambda FLC is defined as involved FLC, and Kappa FLC is defined as non-involved FLC. Then:
  - o Difference between involved and uninvolved = Lambda FLC Kappa FLC.
- If the baseline ratio of (Kappa FLC/Lambda FLC) ≥ 0.26 and ≤ 1.65, then "involved" and "non-involved" FLC cannot be determined (ratio is normal), and calculation of the maximum percent reduction from baseline for the difference between 2 types of Serum FLC will not be possible.

## 7.1.3. Population of Interest

The mITT Population will support the primary efficacy analyses, while the ITT Population will be used for sensitivity analysis of the primary efficacy endpoint. If the mITT and ITT Populations are identical, then only the results associated with the mITT Population will be reported.

# 7.1.4. Strategy for Intercurrent Events

A composite strategy will be followed for participants who are not evaluable or have missing BOR who will be treated as non-responders; i.e., they will be included in the denominator when calculating the percentage.

# 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and based on GSK data standards and statistical principles.

# 7.2. Secondary Efficacy Analyses

### 7.2.1. Endpoints/Variables

# 7.2.1.1. Time to Response (TTR)

TTR is defined as the time interval (in months) from T-cell infusion to initial date of documented confirmed response (PR or better) in the subset of participants who showed a confirmed BOR of PR or better by Investigator assessment per IMWG (2016).

# 7.2.1.2. Duration of Response (DoR)

DoR is defined as the time interval (in months) from initial date of documented confirmed response (PR or better) to the date of confirmed PD or death due to disease under study for participants who showed a confirmed BOR of PR or better IMWG (2016).

Although documentation of responses of PR and better requires a confirmatory measurement, the start time for DoR will be the first date on which response was noted (i.e., the date of "first assessment", as described in Section 7.1.1, Primary Endpoint/Variable: Overall Response Rate (ORR)). Determination of event/censoring for DoR events and associated dates are described in Table 3.

Note that, for participants who receive subsequent anti-cancer therapy, no imputation will be performed for completely missing start dates. However, if the start date of the anti-cancer therapy is partial (i.e., either missing the day but has the month and year available or missing both day and month), then the imputation rules described in Section 14.7.2.1, Handling of Missing and Partial Dates, will be applied.

Table 3 Assignments for Progression/Death and Censoring Dates for DoR Analysis

| Scenario | Date of Event or Censoring | <b>Event or Censored</b> |
|---|---|---|
| No (or inadequate) baseline assessment <sup>[1]</sup> and the participant has not died (if the participant has died, follow the rules for death at the bottom of this table). | Date of T-cell infusion | Censored |
| No post-baseline assessments<br>and the participant has not died<br>(if the participant has died,<br>follow the rules for death at the<br>bottom of this table). | Date of T-cell infusion | Censored |
| New anti-cancer therapy started<br>on or after lymphodepletion and<br>prior to T-cell infusion | Date of T-cell infusion | Censored |
| PD documented at or between scheduled visits. | Date of documented PD <sup>[3]</sup> | Event |

| Scenario | Date of Event or Censoring | <b>Event or Censored</b> |
|---|---|---|
| With post-baseline assessment | Date of last adequate disease | Censored |
| but no PD or death. | assessment <sup>[2]</sup> | |
| New anti-cancer therapy started | Date of last adequate disease | Censored |
| prior to documented PD or | assessment <sup>[2]</sup> on or prior to starting | |
| death <sup>[3]</sup> . | anti-cancer therapy | - |
| Death due to disease under | Date of death | Event |
| study without extended loss to | | |
| follow-up. Death from causes other than | Date of death | C1 |
| disease under study without | Date of death | Censored |
| extended loss to follow-up. | | |
| Death or PD after extended loss | As the schedule of assessments | Censored |
| to follow-up of 2 or more | (Myeloma markers labs) changes | Censored |
| cycles $+ \frac{1}{3}$ 7-day window. | through the course of the protocol | |
| l system in the many will all with | (i.e., starting on Week 1 and then | |
| | every 3 weeks from Week 3 until | |
| | Week 24 and then every 6 weeks | |
| | until Week 72, then every 12 weeks | |
| | until PD), the following rules will be | |
| | used for identifying extended loss to | |
| | follow-up or extended time without | |
| | an adequate assessment (i.e., 2 or | |
| | more missed assessments + window). | |
| | • If death or PD is on or prior to | |
| | Day 45 (= Week 6 + 3-day | |
| | window), then participant status | |
| | will be labelled "extended loss to | |
| | follow-up" if the participant did | |
| | not have an adequate assessment | |
| | during the period of 37 days (= 2 | |
| | weeks + 3 weeks + 1-day window | |
| | + 1-day window) prior to death or | |
| | PD; | |
| | • Else if death or PD is after Day 45 | |
| | (= Week 6 + 3-day window) and | |
| | on or prior to Day 175 (= Week 24 | |
| | + 7-day window), then participant | |
| | status will be labelled "extended | |
| | loss to follow-up" if the | |
| | participant did not have an | |
| | adequate assessment during the | |
| | period of 48 days (= 3 weeks + 3 | |
| | weeks + 3-day window + 3-day | |
| | window) prior to death or PD; | |
| | • Else if death or PD is after Day | |
| | 175 (= Week 24 + 7-day window) | |
| | and on or prior to Day 504 (= | |
| | Week 72 + 7-day window), then | |

208470

| Scenario | Date of Event or Censoring | <b>Event or Censored</b> |
|---|---|---|
| | participant status will be labelled "extended loss to follow-up" if the participant did not have an adequate assessment during the period of 98 days (= 6 weeks + 6 weeks + 7-day window + 7-day window) prior to death or PD; | |
| | • Else if death or PD is after Day 504 (= Week 72 + 7-day window), then participant status will be labelled "extended loss to follow-up" if the participant did not have an adequate assessment during the period of 182 days (= 12 weeks + 12 weeks + 7-day window) prior to death or PD. | |
| | DoR will be censored on the date of last adequate disease assessment prior to PD/death. <sup>[2]</sup> | |

Adequate baseline assessment is defined as a baseline assessment with at least one serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP), or involved FLC result available for analysis.

# 7.2.1.3. Progression Free Survival (PFS)

PFS is defined as the time interval (in months) between the date of T-cell infusion and the initial assessment date of confirmed PD as assessed by the investigator per IMWG (2016) or date of death due to any cause. Determination of dates of PFS events and dates for censoring are described in Table 4.

Table 4 Assignments for Progression and Censoring Dates for PFS Analysis

| Scenario | Date of Event (Progression/Death)<br>or Censoring | Event<br>(Progression/Death)<br>Or Censored |
|---|---|---|
| No (or inadequate) baseline assessment <sup>[1]</sup> and the participant has not died (if the participant has died, follow the rules for death at the bottom of this table). | Date of T-cell infusion | Censored |
| No post-baseline assessments and the participant has not | Date of T-cell infusion | Censored |

<sup>&</sup>lt;sup>2</sup> Adequate disease assessment is defined as a disease assessment with Investigator-assessed response of sCR, CR, VGPR, PR, MR, or SD per IMWG (2016). The date of response will be recorded on the Disease Assessment eCRF.

<sup>&</sup>lt;sup>3</sup> If PD (or death) and new anti-cancer therapy occur on the same day, the assumption will be made that PD (or death) was documented first (i.e., PD would equal the outcome and the relevant date would be the date of documented PD). If anti-cancer therapy is started prior to any adequate disease assessments (but after lymphodepleting chemotherapy), the censoring date will equal the date of T-cell infusion.

| Scenario | Date of Event (Progression/Death) | Event |
|---|---|---|
| | or Censoring | (Progression/Death) Or Censored |
| died (if the participant has died, follow the rules for death at the bottom of this table). | | |
| PD documented between scheduled visits, without extended loss to follow-up. | Date of documented PD <sup>[3]</sup> | Event |
| With post-baseline assessment but no documented PD or death. | Date of last adequate disease assessment <sup>[2]</sup> | Censored |
| No adequate post-baseline assessment before start of new anti-cancer therapy. | Date of T-cell infusion | Censored |
| With adequate post-baseline assessment and new anti-cancer therapy started prior to documented PD or death <sup>[3]</sup> . | Date of last adequate disease assessment <sup>[2]</sup> on or prior to starting anti-cancer therapy | Censored |
| Death before first scheduled assessment, or death at baseline without adequate baseline assessment, or death following a post-baseline assessment (i.e., "between assessments") without extended loss to follow-up. | Date of death | Event |
| Death or PD after extended loss to follow-up or time without adequate disease assessment of 2 or more cycles + 1/3/7-day window | As the schedule of assessments (Myeloma markers labs) changes through the course of the protocol (i.e., starting on Week 1 and then every 3 weeks starting from Week 3 until Week 24 and then every 6 weeks until Week 72, then every 12 weeks until PD), the following rules will be used for identifying extended loss to follow-up or extended time without an adequate assessment (i.e., 2 or more missed assessments + window). • If death or PD is after Day 45 (= Week 6 + 3-day window) and on or prior to Day 175 (= Week 24 + 7-day window), then participant status will be labelled "extended loss to follow-up" if the participant did not have an adequate assessment during the period of 48 days (= 3 weeks + 3 weeks + 3-day) | Censored |

208470

| Scenario | Date of Event (Progression/Death) or Censoring | Event<br>(Progression/Death)<br>Or Censored |
|---|---|---|
| | window + 3-day window) prior to death or PD; | |
| | • Else if death or PD is after Day 175 (= Week 24 + 7-day window) and on or prior to Day 504 (= Week 72 + 7-day window), then participant status will be labelled "extended loss to follow-up" if the participant did not have an adequate assessment during the period of 98 days (= 6 weeks + 6 weeks + 7-day window) prior to death or PD; | |
| | • Else if death or PD is after Day 504 (Week 72 + 7-day window), then participant status will be labelled "extended loss to follow-up" if the participant did not have an adequate assessment during the period of 182 days (12 weeks + 12 weeks + 7-day window + 7-day window) prior to death or PD. PFS will be censored on the date of last adequate disease assessment (or T-cell infusion, if no adequate disease assessment) prior to PD/death. <sup>[2]</sup> | |

Adequate baseline assessment is defined as a baseline assessment with at least one serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP), or involved FLC result available for analysis.

## 7.2.2. Summary Measure

#### 7.2.2.1. Time to Response (TTR)

Time to response for each participant with a confirmed response (PR or better) will be listed in months. Details are provided in Appendix 12.

<sup>&</sup>lt;sup>2</sup> Adequate disease assessment is defined as a disease assessment with Investigator-assessed response of sCR, CR, VGPR, PR, MR, or SD per IMWG (2016). The date of response will be recorded on the Disease Assessment eCRF.

<sup>&</sup>lt;sup>3</sup> If PD (or death) and new anti-cancer therapy occur on the same day, the assumption will be made that PD (or death) was documented first (i.e., PD would equal the outcome and the relevant date would be the date of documented PD). If anti-cancer therapy is started prior to any adequate disease assessments (but after starting lymphodepleting chemotherapy), the censoring date will equal the date of T-cell infusion.

#### 7.2.2.2. Duration of Response

Duration of response for each participant with a confirmed response (PR or better) will be listed in months. Details are provided in Appendix 12.

#### 7.2.2.3. Progression Free Survival

PFS will be summarized using Kaplan-Meier curves. Median PFS, first and third quartiles and 95% CI, will be estimated using the Brookmeyer-Crowley method [Brookmeyer, 1982]. A listing of PFS times and associated details will also be provided. Details of the planned displays are provided in Appendix 12.

#### 7.2.3. Population of Interest

Secondary efficacy analyses will be based on the mITT Population.

## 7.2.4. Statistical Analyses / Methods

Details of the planned displays will be provided in Appendix 12: List of Data Displays and are based on GSK data standards and statistical principles. Unless otherwise specified, endpoints / variables defined above in Section 7.2.2 will be summarized by arm using descriptive statistics, graphically presented (as appropriate), and listed.

# 7.3. Exploratory Efficacy Analyses

MRD will not be analysed at part of this RAP.

#### 7.3.1. Endpoints/Variables

#### 7.3.1.1. Overall Survival (OS)

OS is defined as the time interval (in months) from the date of T-cell infusion to the date of death due to any cause.

Survival outcomes for subjects who have not died by the point of analysis will be censored on the date of last known contact with the participant.

## 7.3.2. Summary Measure

OS for each participant will be listed in months.

#### 7.3.3. Population of Interest

The exploratory efficacy analysis will be based on the mITT Population.

#### 7.3.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and are based on GSK data standards and statistical principles. Unless otherwise specified,
# 208470l Statistical Analysis Plan RAP 23 Apr 2021 | TMF-13337917 | 1.0

# CONFIDENTIAL

208470

endpoints / variables defined in Section 7.3.1 will be summarized using descriptive statistics, graphically presented (if appropriate), and listed.

208470

## 8. SAFETY ANALYSES

The safety analyses will be based on the Intent-to-Treat population except for displays that are treatment dependent where the modified Intent-to-Treat population will be used, as detailed in Appendix 12.

Unless otherwise specified, summaries will include descriptive statistics by treatment arm, as well as overall (across treatment arms).

# 8.1. Adverse Events Analyses

Analysis of AEs, including all AEs, serious AEs (SAEs), and other significant AEs, will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 12: List of Data Displays.

AEs will be graded according to National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 4.03 unless otherwise specified in the protocol. For instance, the grading of AE-related Cytokine Release Syndrome (CRS) will be performed using modified NCI-CTCAE guidance developed by Lee (2019, Section 13); see protocol Table 5 and Section 8.5. For the grading of Graft versus Host Disease (GVHD) associated AEs, see protocol Section 8.6.2. AEs will be coded to the level of Preferred Term (PT) using the latest version of the Medical Dictionary for Regulatory Affairs (MedDRA).

In the eCRF for this study Adverse Events for which the grade changes over the course of the event are entered as multiple records, one record per grade. (If multiple grades are experienced on the same day then the highest grade for that day is reported.) Similarly, events where other attributes such as relatedness change over the course of the event will also be entered as multiple records. For analyses requiring summaries of numbers or characteristics of individual events, these multiple sequential segments will be collapsed back into a single event record prior to analysis using the algorithm detailed in Appendix 15

AEs related to study treatment, SAEs, SAEs related to any study treatment, fatal AEs, and fatal AEs related to any study treatment will be summarized.

Tables will summarize all AEs for the ITT population and Treatment Emergent AEs for the MITT population.

A summary of common non-serious AEs that occurred strictly in  $\geq 5\%$  of participants will be provided, without rounding of the percentage to overcome the 5% threshold (e.g., events with 4.9% incidence rate will not be included). This summary will display the number and percentage of participants, while a separate summary will present the total numbers of occurrences of the common non-serious AEs. Both summary tables will be displayed by MedDRA System Organ Class (SOC) and PT.

The relationship between MedDRA SOC, PT, and Verbatim Text will be listed.

208470

A summary of number and percentage of participants with any AEs by maximum grade will be produced. AEs will be sorted by combined PT in descending order of total incidence. The summary will use the following algorithms for counting the participant:

- **Preferred term row**: Participants experiencing the same AE preferred term several times with different grades will only be counted once with the maximum grade.
- **Any event row**: Each participant with at least one AE will be counted only once at the maximum grade no matter how many events they have.

In addition, the frequency and percentage of AEs (all grades) will be summarized and displayed in 2 ways: 1) in descending order of total incidence by combined PT only and 2) in descending order of total incidence by SOC and PT. In the SOC row, the number of participants with multiple events under the same SOC label will be counted once.

A study treatment-related AE is defined as an AE for which the investigator classifies the relationship to lymphodepleting chemotherapy, T-cell infusion, and/or pembrolizumab as "Yes", which includes "Definitely Related", "Probably Related", and "Possibly Related". Summary of study treatment related AEs by combined PT and maximum grade will also be provided separately for relatedness to each study treatment. A worst-case scenario approach will be taken to handle missing relatedness data (i.e., the summary table will include events with the relationship to study treatment as 'Yes' or missing).

In addition to the summaries and listings described above, listings will be provided for all AEs, AEs leading to pembrolizumab dose interruption (in Arm 2), AEs leading to pembrolizumab dose reduction (in Arm 2), AEs leading to pembrolizumab dose discontinuation (in Arm 2), delayed AEs as adjudicated by GSK (provided from external data source), and participant IDs per individual AE.

Tables that summarize AEs by SOC and PT will use MedDRA preferred terms, as well as any adverse event tables required for disclosure. This will be detailed in the programming notes in Appendix 12: List of Data Displays. Most other AE tables will summarize AEs by using the combined terms defined in Appendix 14: Combined Preferred Terms, as detailed in the programming notes in Appendix 12: List of Data Displays.

In the event that a participant has withdrawn consent, no data after the withdrawal of consent date from this participant including death should appear in the database, which should be part of the data cleaning process. All deaths will be summarised based on the number and percentage of participants. This summary will classify participants by time of death relative to the date of T-cell infusion (>30 days or ≤30 days) and primary cause of death (disease under study, treatment related toxicity, or other). A supportive listing will be generated to provide participant-specific details on participants who died.

AEs deemed serious are those events leading to death, life-threatening circumstance, or new/prolonged hospitalization or, given appropriate medical judgement, requires medical or surgical intervention to prevent one or more of the aforementioned outcomes (see protocol Section 9.3 for more detail). Separate summaries will be provided for AEs (and SAEs) related to study treatments: one for lymphodepleting chemotherapy-related (S)AEs, one for T-cell infusion-related (S)AEs, and one for all study treatment related

208470

(S)AEs. Summaries of fatal AEs, and fatal AEs related to any study treatment will be produced. Fatal AEs will only be summarized if there are at least 5 participants with fatal AEs.

SAEs will be included in the listing of all AEs, but also separate supportive listings with participant-level details will be generated for:

- Non-fatal SAEs
- Reasons for considering AE as serious

A summary of total incidence and frequency and percentage of grade 3, 4, and 5 events will be presented by study arm and total for the following: all AEs, all treatment emergent AEs, all study-treatment related AEs, all T-cell related AEs, all lymphodepletion related AEs, all serious AEs, and all study-treatment related, T-cell related, and lymphodepletion related serious AEs.

A plot of study duration including study days of any SAE, death, progression, and response will be produced.

# 8.2. Adverse Events of Special Interest (AESI) Analyses

### AESIs include:

- Cytokine Release Syndrome
- Haematopoietic cytopenias (including pancytopenia and aplastic anaemia)
- Graft versus Host Disease (GvHD)
- Immune Effector-Cell Associated Neurotoxicity Syndrome (ICANS)
- Guillain-Barre Syndrome (GBS)

A focused list of MedDRA terms based on clinical review will be used to identify each type of event. In addition, all potential haematopoietic cytopenias will be identified using a comprehensive list of MedDRA terms. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting, and emerging data from on-going studies may highlight additional AEs of special interest (AESIs). Therefore, the list of terms to be used for each event of interest and the specific events of interest will be based on the SRT agreements in place at the time of reporting. Due to expected small numbers, Gullian-Barre Syndrome, Immune Effector-Cell Associated Neurotoxicity Syndrome, and Graft versus Host Disease will only be displayed in listings. Details of the planned displays are provided in Appendix 12: List of Data Displays.

AESI tables will be reported for the mITT population.

The number and percentage of participants with these events will be summarized by categories of AESI, combined preferred term, and grade in one table using both the comprehensive list and focused list. All additional AESI tables described below will be summarized using the focused list and additional Haematopoietic cytopenia AESI tables

208470

will also be summarized by cell line, using the specific neutropenia, thrombocytopenia, and anemia preferred terms in the focused list.

Listings of AESIs will be produced for each AESI category using the focused list, which will include leukapheresis date, lymphodepletion start date, T cell infusion date, AE start date, AE end date, SAE code, grade, relationship to study treatment and outcome of event. An additional listing of cytopenias identified in the comprehensive list will also be provided.

The summary of event characteristics for each category of AESI will also be provided, including number of participants with any event, number of events, number of participants with any event that is related to study treatment, the outcome of the event, maximum grade and the action taken for the event. The percentage will be calculated in 2 ways, one with number of participants with event as the denominator and the other with total number of participants as the denominator. The worst-case approach will be applied at participant level for the event outcome and maximum grade, i.e. a participant will only be counted once as the worst case from all the events experienced by the participant. For action taken to an event, participant will be counted once under each action, e.g. if a participant has an event leading to both study treatment discontinuation and dose reduction, the participant will be counted once under both actions.

A summary of onset and duration of the first occurrence of all AESIs will be created for each AESI separately, and for Haematopietic cytopenias this will include an overall analysis of events in the focused list of PTs for this AESI as well as separate analyses for cell lines describing events of Neutropenia, Anemia, and Thrombocytopenia. A summary of onset and duration of the last occurrence of focused list Haematopoietic cytopenias will also be created. In addition, a summary of time to resolution will be created for each AESI separately. The time to resolution displays summarize participants with an AESI occurring before study day 30. Among all AESIs occurring before study day 30, the worst-case study day of resolution will be summarized. Additionally, the worst-case AESI duration of all recurrent AESIs will be summarized. Recurrent AESI is defined as additional occurrences of AESIs after day 30, after initial occurrence and before study day 30. Duration is defined as AESI end date – AESI start date + 1.

Characteristics, Onset and Duration, and Time to Resolution summaries will not be created if there are 0 or 1 AESI in total.

# 8.2.1. Cytokine Release Syndrome (CRS) and Graft versus Host Disease (GvHD)

Refer to protocol Section 8.5 and Section 8.6 for the definitions and the grading of CRS and GvHD. The listing of CRS AESIs will also include time from infusion to first CRS (days) and time from infusion to max CRS (days). Listings of symptoms, medications and procedures related to CRS and GvHD will be produced separately. The mock-up shells are in Appendix 13: Example Mock Shells for Data Displays.

# 8.3. Clinical Laboratory Analyses

Laboratory evaluations including chemistry, hematology, and other laboratory tests, including biomarker tests, will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12: List of Data Displays.

The laboratory assessments to be conducted for monitoring participant safety are listed in Table 5, List of Clinical Laboratory Tests.

Table 5 List of Clinical Laboratory Tests

| Clinical Chemistry | Hematology |
|---|---|
| Total Calcium | Red blood cell count |
| Calcium corrected for Albumin | Hemoglobin |
| Phosphorus | Hematocrit |
| Magnesium | Mean cell volume |
| Albumin | Mean corpuscular hemoglobin |
| Bilirubin | Mean corpuscular hemoglobin concentration |
| Alanine aminotransferase | Platelet count |
| Aspartate aminotransferase | White blood cell count |
| Alkaline phosphatase | White blood cell differential absolute counts of |
| Lactate dehydrogenase | lymphocytes, monocytes, and neutrophils |
| Sodium | White blood cell differential percentages of lymphocytes, monocytes, and neutrophils |
| Potassium | lymphocytes, monecytes, and neutrophilis |
| Bicarbonate | |
| Creatinine* | |
| Chloride | |
| Glucose | |
| BUN or Urea | |
| Uric Acid | |
| C-reactive protein | |
| * In participants ≥65 years, add GFR | |

208470

| Other Clinical Lab tests | |
|---|---|
| Urinalysis: | Immunology: |
| Glucose | HIV 1+2 antibody |
| Ketones | Hepatitis B surface antigen |
| Specific gravity | Hepatitis B core antibody – if positive, test for |
| Protein | HBV DNA |
| Blood | Hepatitis C antibody – if positive, test for HCV |
| Microscopy | RNA |
| Bilirubin | HTLV 1+2 IgG |
| pH | CMV IgG |
| | EBV (EBNA) |
| Coagulation: | Syphilis (RPR) |
| Congulation | CMV DNA PCR – peripheral blood for |
| Prothrombin time or International | detection of reactivation. |
| Normalized Ratio | |
| Activated partial thromboplastin time | |
| | Pregnancy: |
| Endocrinology: | Serum beta-HCG or urine test |
| Thyroid stimulating hormone | |
| Myeloma markers: | |
| SPEP | |
| UPEP | |
| IgG | |
| IgM | |
| IgA | |
| Serum free Kappa chain | |
| Serum free Lambda chain | |
| Kappa/Lambda ratio determination | |
| Beta-2 microglobulin | |
| Serum M-protein | |
| Serum Immunofixation | |

Summaries of worst-case grade increase from baseline grade at Week 4, Week 15, and across all post-baseline visits will be provided for all the lab tests that are gradable by NCI-CTCAE v4.03. The worst grade will be derived based on all post baseline records including unscheduled visits. These summaries will display the number and percentage of participants with a maximum post-baseline grade increasing from their baseline grade. Missing baseline grade will be assumed as grade 0. For laboratory tests that are graded for both low and high values, summaries will be done separately and labeled by direction, e.g. sodium will be summarized as hyponatremia and hypernatremia.

For lab tests that are not gradable by NCI-CTCAE v4.03, summaries of worst-case changes from baseline with respect to normal range will be generated. Decreases to low,

208470

changes to normal or no changes from baseline, and increases to high will be summarized at each scheduled visit as well as for the worst-case post-baseline. If a participant has a decrease to low and an increase to high during the same time interval, then the participant is counted in both the "Decrease to Low" categories and the "Increase to High" categories. In addition, the summary will include worst-case changes from baseline with respect to normal range for worst cases.

Separate summary tables for hematology, chemistry, and other laboratory tests will be produced. Summary of the change from baseline for hematology, chemistry, and other lab tests will be provided by visit using n, mean, median, standard deviation, minimum, and maximum. A plot of each subject's laboratory data over time will be created for the following hematologic tests: neutrophils, lymphocytes, platelets, and hemoglobin. Additionally, all laboratory values will be provided in a listing.

Detailed derivation of baseline assessment is specified in Section 5.2, Baseline Definitions. Unless otherwise specified, the denominator used in calculating percentage at each scheduled visit will equal the number of participants with non-missing values at the particular visit.

# 8.3.1. Analyses of Liver Function Tests (LFT)

Listings of hepatobiliary laboratory events including possible Hy's law cases will be provided in addition to what has been described above, including listings of liver monitoring and stopping events as well as a listing of subjects meeting hepatobiliary laboratory criteria post-baseline.

Possible Hy's law cases will be defined as any event of either: (a) alanine aminotransferase (ALT)  $\geq$ 3 × the upper limit of normal (ULN) and bilirubin  $\geq$ 2 × ULN (>35% direct bilirubin) or (b) ALT  $\geq$ 3 × ULN and INR >1.5, if INR is measured. Total bilirubin  $\geq$ 2 × ULN can be within 28 days following the ALT elevation and, if direct bilirubin is available on the same day, it must be  $\geq$ 35% of total bilirubin. Note that INR measurement is not required, and the threshold value stated will not apply to participants receiving anticoagulants.

A scatter plot of maximum total bilirubin versus maximum ALT will be generated. Also, a scatter plot of maximum vs baseline for ALT will be produced.

# 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results, including ECGs and vital signs, will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 12: List of Data Displays.

### 8.4.1. Performance Status

Eastern Cooperative Oncology Group (ECOG) performance status at baseline and at the participant's last assessment will be summarized. A summary of change from baseline by scheduled visits will also be produced, including the worst-case and best-case post-

208470

baseline changes during the study (improved, no change, deteriorated). Summaries will use frequency and percentage of participants at each planned assessment time. A supportive listing will also be provided.

### 8.4.2. ECG

A summary of the number and percentage of participants who had normal and abnormal (clinically significant and not clinically significant) ECG findings will be displayed by scheduled visits as well as for the worst-case post-baseline. The worst case will be chosen from all available ECG findings, including scheduled and unscheduled visits.

A summary of change from baseline in ECG values will be produced.

A summary of increases in QTc comparing the baseline value to worst-case post baseline value will be provided. The worst-case post baseline row is used to summarize the participants' overall worst-case shifts post baseline. The determination of the worst-case post baseline takes into account both planned and unscheduled assessments. In addition, the summary also includes a comparison of the worst-case shifts by planned time intervals.

Similarly, the amount of increase from baseline in QTc values will also be summarized. Participants with missing baseline values will be excluded from this summary.

Summaries of QTc values will incorporate corrections based on Friderica's or Bazett's formula separately (with values referred to as QTcF and QTcB, respectively).

Listings of abnormal ECG findings and a listing of ECG values will be provided.

A figure plotting QTc shift from baseline to worst-case post baseline will be produced, with separate plots for the 2 correction methods (QTcF and QTcB). Plots within the figure will have reference lines at 480 and 500 msec for both the ordinate and abscissa axes. There will be diagonal reference lines at equality (i.e., a 45-degree line), at equality plus 30 msec, and at equality plus 60 msec.

### 8.4.3. Pregnancies

Pregnancy (or pregnancy of a male participant's partner) is not considered an AE/SAE unless there is reason to believe that the pregnancy may be the result of failure of the contraceptive being used due to interaction with the study drug. However, the investigator shall report all pregnancies immediately to the Sponsor. If participants or participants' partner become pregnant while on the study, the information will be included in the narratives and no separate table or listing will be produced.

### 8.4.4. Vital Signs

A summary of change from baseline in vital signs will be provided. Also, a summary of worst-case vital signs results by Potential Clinical Importance (PCI) criteria post-baseline relative to baseline will be generated (see Appendix 8: Values of Potential Clinical Importance).

A listing of vital signs with values of PCI will be provided.

# 8.4.5. Replication Competent Lentivirus (RCL) and Persistence of NY-ESO-1<sup>c259</sup>T

The proportion of participants who are RCL positive will be summarized. RCL is reported as "Negative" if copies of VSV-G are <50 copies/ug DNA.

RCL results will also be presented in a data listing.

The proportion of patients showing >1% gene marked peripheral blood mononuclear cells (PBMCs) one-year post-treatment will be summarized if data warrant.

For any patient who has greater than 1% gene marked PBMCs at 1 year or beyond post-infusion, integration site analysis will be performed on PBMCs to assess clonality and possible insertional oncogenesis. A summary of the number of subjects with any number of clones with >7% abundance will be summarized if data warrant. A supporting listing will be provided. Two diversity indices, Shannon diversity index and Gini index, will be reported in the data listing. These indices can help summarize the composition of a population of clones. Shannon diversity is a measurement that represents the uncertainty about the identity of a single species within the population [Shannon, 1948, Section 13]. The Gini index can help detect the similarity in abundance of different clones across the population [Gini, 1914, Section 13]

Further details of the handling of persistence data and its analysis as a biomarker are given in Section 9.1.

### 8.4.6. COVID-19

A listing of all COVID-19 assessments, including test date and result, along with symptom assessments will be provided.

### 9. PHARMACOKINETIC ANALYSES

# 9.1. Primary Pharmacokinetic Analyses

# 9.1.1. Endpoint / Variables

Evaluation of persistence of NY-ESO-1<sup>c259</sup>T cells over time is a secondary objective.

### 9.1.1.1. Drug Concentration Measures

Spider plots will be used to graphically summarize persistence over time for each participant by responders and non-responders. Spider plots of Bone Marrow Mononuclear Cell (BMMC) persistence data will also be produced if data is available.

### 9.1.1.2. Derived Pharmacokinetic Parameters

The PK parameters presented in the table below will be derived during programming. This will be the responsibility of the Statistics and Programming group at PAREXEL under the direction of the Clinical Pharmacology Modeling and Simulation (CPMS) Department at GSK.

Peak expansion during the study (Cmax), time to peak expansion (Tmax), and as data permit,  $AUC_{(0-28)}$  will be summarized overall and for responders and non-responders using descriptive statistics and dot plots.

The area under the plasma concentration-time curve to day 28 (AUC<sub>(0-28)</sub>) will be determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. PK samples intended for day 28 will be treated as collected on that day provided they are collected within 4 days of day 28.

# 9.1.2. Summary Measure

For each of these parameters, except Tmax, the following summary statistics will be calculated: n, median, minimum, maximum, arithmetic mean, 95% confidence interval for the arithmetic mean, standard deviation, coefficient of variation (CV) =  $100*(sqrt(exp(SD^2) - 1)))$  [NOTE: SD = SD of log transformed data]), geometric mean, 95% confidence interval for the geometric mean and standard deviation of logarithmically transformed data. Data will be summarized by treatment arm and overall, and by type of persistence if BMMC persistence data is available.

For Tmax, calculations will include median, maximum, minimum, arithmetic mean, 95% confidence interval, and standard deviation. Data will be summarized by treatment arm and overall.

A listing of persistence will be provided and will include coefficient of variation, number of positive replicates, copies/cell, copies/ $\mu$ g DNA, percent gene marked cells of PBMCs (%), interpretive result, duration of detectible persistence, time to loss of 25%/50%/75% peak expansion, and AUC<sub>(0-28)</sub>. An identical persistence listing will be created for BMMC data.

Time to loss of 25% of peak expansion will be calculated as the time since T-cell infusion corresponding to observing at least 25% loss of peak expansion. If time to 25% loss of peak expansion is not observed, the last observed time will be reported with a "+". The same procedure will be followed for 50% and 75%.

The following calculations will be performed:

copies/cell is calculated with the following formula:

copies/cell=(copies/µg) x (0.0000063 µg gDNA/cell)

Percent gene-marked cells of peripheral blood mononuclear cells (PBMCs) = (copies/cell) x 100

The final reported result of copies/µg gDNA is calculated as follows:

copies/µg DNA=copies per well/µg gDNA per well

For persistence value below LLOQ, the following rules will be applied:

| Reported Copies<br>per cell Result | Reported Copies<br>per ug gDNA<br>Result | Reported Result | Set Value for<br>Copies per cell | Set Value for<br>Copies per ug<br>gDNA |
|---|---|---|---|---|
| <0.0003 | <50.0 | Negative | 0 | 0 |
| <0.0003 | <50.0 | Detectable,<br><lloq< td=""><td>0.0003</td><td>50</td></lloq<> | 0.0003 | 50 |

Note, sometimes values for copies per cell and copies per ug DNA might be different than above as it depends on the input of DNA, but rule would be the same:

- If interpretive reported result is negative, then set values to 0.
- If interpretive reported result is "Detectable, <LLOQ", set values to LLOQ (If <XXX, set at XXX)

The unit for persistence will be "Copies/ug of gDNA"

Duration of detectable persistence is defined as time from T-cell infusion until persistence is no longer detectable. Persistence above the assay limit of detection but below the lower limit of quantitation is considered for the duration determination, i.e. the time window from infusion until the first instance persistence falls below the detection limit and the interpretive reported result is "Negative." If persistence for a given participant remains detectable ("Positive" or "Detectable, LLOQ") at their last sample collection timepoint, the last observed time is reported and considered as right-censored with a "+" appended to the numerical result. Note, transduced T-cells frequently persist beyond the follow-up period, and hence, the reported duration is directly influenced by length of time the participant is on-study

### 9.1.3. Population of Interest

All analyses of persistence will be based on the mITT population, unless otherwise specified.

# 10. BIOMARKER ANALYSES

# 10.1. Biomarker Analyses

# 10.1.1. Endpoint / Variables

Anti-NYESO antibody formation will be reported if data warrant.

# 10.1.2. Summary Measure

## 10.1.2.1. Anti-NYESO-1 Antibody Formation

The anti-NY-ESO-1 antibody results, including titers, will be reported for all participants in a data listing. Additionally, the overall incidence of participants with all negative or confirmed positive results at baseline and any post-treatment time point will be summarized if data warrant.

# 10.1.3. Population of Interest

Biomarker analyses will be based on the mITT Population, unless otherwise specified.

# 10.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and are based on GSK data standards and statistical principles.

# 11. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

Not applicable.

# 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

Not applicable.

208470

# 13. REFERENCES

Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics, 1982; 38:29-41.

Gini C. Sulla misura della concentrazione e della variabilita dei caratteri. Transactions of the Real Istituto Veneto di Scienze. 1914; LIII:1203Appendices

Kumar S, Pariva B, Anderson KC, et al. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. The Lancet. 2016;17;e328-e346.

Lee DW, Santomasso BD, Locke FL, et al. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol. Blood Marrow Transplant. 2019;25:625-638.

Lee JJ, Liu DD. A predictive probability design for phase II cancer clinical trials. Clin Trials. 2008;5(2):93-106.

Shannon, C. A mathematical theory of communication. Bell Syst. Tech. J. 1948;27:379–423, 623–656.

208470

# 14. APPENDICES

# 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Specification document.

208470

# 14.2. Appendix 2: Schedule of Activities

# 14.2.1. Protocol Defined Schedule of Events

| | | | Treatment Phas | se | | | | | | | | | | | | | | | | | | DC of | Comple- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Phase<br>/<br>Eligit<br>Phase | ility | Leukapheresis | Baseline ≤7 days prior to chemo | Lym<br>Che | nphoc<br>moth | deple<br>erap | ting<br>y <sup>b</sup> | | T-cell<br>infu-<br>sion | | | | | | | | | | | | Pem-<br>broli-<br>zumab<br>Tx <sup>c</sup> | tion of<br>Treatment<br>Phase or<br>WDd |
| Study Day | Scrn | Elig | | D -14 to<br>D -8 | D -<br>8 | D-7 | D- | D -<br>5 | D -<br>4 | D 1 | D2 | D3 | D4 | D5 | Wk<br>1 | Wk<br>2 | Wk<br>3 | Wk<br>4 | Wk<br>6 | Wk<br>15 | Wk 24<br>&<br>Q12wks | | |
| Window | | | | | | | | | | | | | | | ±1D | ±1D | ±1D | ±3D | ±3D | ±3D | ±7D | | |
| Informed consent <sup>a</sup> | Х | Х | | | | | | | | | | | | | | | | | | | | | |
| Demographics | Х | | | | | | | | | | | | | | | | | | | | | | |
| HLA-genotyping | Х | | | | | | | | | | | | | | | | | | | | | | |
| NY-ESO-1 and<br>LAGE-1a levels<br>on BM aspirate | Х | | | | | | | | | | | | | | | | | | | | | | |
| Inclusions/<br>Exclusions | | Х | | Х | | | | | | | | | | | | | | | | | | | |
| Baseline characteristics <sup>e</sup> | | | | Х | | | | | | | | | | | | | | | | | | | |
| Medical History <sup>f</sup> | | Х | | | | | | | | | | | | | | | | | | | | | |
| Physical Exam <sup>9</sup> | | Х | | Х | | | | | | | | | | | | | | | | | Х | | |
| Prior/Concomitant medicationh | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | х | X | х |

| | Scree | ninga | Treatment Phas | se | | | | | | | | | | | | | | | | | | DC of | Comple- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Phase<br>/<br>Eligib<br>Phase | ility | Leukapheresis | Baseline ≤7 days prior to chemo | | | deple<br>erap | | | T-cell<br>infu-<br>sion | | | | | | | | | | | | Pem-<br>broli-<br>zumab<br>Tx <sup>c</sup> | tion of<br>Treatment<br>Phase or<br>WDd |
| Study Day | Scrn | Elig | | D -14 to<br>D -8 | D -<br>8 | D-7 | D -<br>6 | D -<br>5 | D -<br>4 | D 1 | D2 | D3 | D4 | D5 | Wk<br>1 | Wk<br>2 | Wk<br>3 | Wk<br>4 | Wk<br>6 | Wk<br>15 | Wk 24<br>&<br>Q12wks | | |
| Window | | | | | | | | | | | | | | | ±1D | ±1D | ±1D | ±3D | ±3D | ±3D | ±7D | | |
| ECOG PS | | Χ | | Х | | | | | | Χ | | | | | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Χ |
| Vital signs /<br>Weight | | Х | | Х | | | | | | Xi | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х | Х | Х |
| Pulse oximetry | | Χ | | Х | | | | | | | | | | | | | | | | | | | |
| ECG | | <b>χ</b> j | | Х <sup>j</sup> | | | | | | Х | | | Χ | | Χ | | | | | | | | |
| Echo / MUGA | | Xa,k | | | | | | | | | | | | | | | | | | | | | |
| Chest X-ray<br>(if indicated) | | Х | | | | | | | | | | | | | | | | | | | | | |
| Hematology | | Χ | | Х | Х | Х | Х | Х | Х | Х | Χ | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Clinical Chemistry | | Χ | | Χ | Х | Х | Х | Х | Х | Х | Χ | Χ | Χ | Χ | Χ | Х | Х | Χ | Χ | Х | Х | Х | Х |
| Coagulation tests | | Χ | | Χ | | | | | | | | | | | | | | | | | | | |
| Pregnancy test <sup>m</sup> | | Χ | | Χ | | | | | | | | | | | | | | | | | | | |
| Urinalysis <sup>l</sup> | | Χ | | Χ | | | | | | | | | | | | | | | | | | | |
| Infectious<br>Disease screen <sup>n</sup> | | X | | | | | | | | | | | | | | | | | | | | | |
| CMV PCRº | | | | Х | | | | | | Х | | | | | Χ | | | Х | Χ | | | | |
| Thyroid Function<br>Testsl | | | | Х | | | | | | Х | | | | | | | | | X then Q6wks (Arm 2 only) | | | | |

| | Scree | ninga | Treatment Phas | se | | | | | | | | | | | | | | | | | | DC of | Comple- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Phase<br>/<br>Eligib<br>Phase | ility | Leukapheresis | Baseline<br>≤7 days<br>prior to<br>chemo | | nphoo | | | | T-cell infu-sion | | | | | | | | | | | | Pem-<br>broli-<br>zumab<br>Tx <sup>c</sup> | tion of<br>Treatment<br>Phase or<br>WD <sup>d</sup> |
| Study Day | Scrn | Elig | | D -14 to<br>D -8 | D -<br>8 | D-7 | D -<br>6 | D -<br>5 | D -<br>4 | D 1 | D2 | D3 | D4 | D5 | Wk<br>1 | Wk<br>2 | Wk<br>3 | Wk<br>4 | Wk<br>6 | Wk<br>15 | Wk 24<br>&<br>Q12wks | | |
| Window | | | | | | | | | | | | | | | ±1D | ±1D | ±1D | ±3D | ±3D | ±3D | ±7D | | |
| C-Reactive<br>Protein <sup>p</sup> | | | | Х | | | | | | Х | | | | Χ | | | Х | | Х | | | | |
| Uric acid | | | | Χ | | | | | | Х | | | | | | | | | | | | | |
| GFR or 24h urine creatinine <sup>q</sup> | | Х | | X | | | | | | | | | | | | | | | | | | | |
| Adverse Events <sup>r</sup> | | Х | Х | Χ | Х | Х | Χ | Х | Х | Х | Х | Х | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Vector Copies<br>(Persistence for<br>safety) <sup>s</sup> | | | | | | | | | | х | | | | | | | | | | Х | Χs | | |
| VSV-G DNA<br>(RCL) for safety <sup>s</sup> | | | | | | | | | | Х | | | | | | | | | | Х | Xs | | |
| Leukapheresis, L | ympho | deple | ting Chemothera | ару | l | | | ı | ı | | l | | | | | 1 | 1 | | 1 | ı | I | | I |
| Leukapheresis <sup>t</sup> | | | Х | | | | | | | | | | | | | | | | | | | | |
| Fludarabine | | | | | Χ | Х | Χ | Х | | | | | | | | | | | | | | | |
| Cyclophospha-<br>mide | | | | | | Х | Х | Х | | | | | | | | | | | | | | | |
| G-CSF <sup>u</sup> | | | | | | | | | Х | | | | | | | | | | | | | | |

| | | | Treatment Phas | | | | | | | | | • | • | • | | | | | | | | DC of | Comple- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Phase<br>/<br>Eligib<br>Phase | ility | Leukapheresis | Baseline<br>≤7 days<br>prior to<br>chemo | | iphoo<br>moth | | | | T-cell<br>infu-<br>sion | | | | | | | | | | | | Pem-<br>broli-<br>zumab<br>Tx <sup>c</sup> | tion of<br>Treatment<br>Phase or<br>WDd |
| Study Day | Scrn | Elig | | D -14 to<br>D -8 | D -<br>8 | D-7 | D -<br>6 | D -<br>5 | D -<br>4 | D 1 | D2 | D3 | D4 | D5 | Wk<br>1 | Wk<br>2 | Wk<br>3 | Wk<br>4 | Wk<br>6 | Wk<br>15 | Wk 24<br>&<br>Q12wks | | |
| Window | | | | | | | | | | | | | | | | ±1D | ±1D | | ±3D | ±3D | ±7D | | |
| Administration of | Inves | tigatio | nal Products | | | | | | 1 | | | | | | | | | ı | | ı | | | |
| NY-ESO-1c259T infusion | | | | | | | | | | X | | | | | | | | | | | | | |
| Pembrolizumab<br>(Arm 2 only) <sup>v</sup> | | | | | | | | | | | | | | | | | X t | X then Q3wks up to Wk108 | | | | | |
| Multiple Myeloma | Disea | se ass | sessments | | | 1 | 1 | | | | | | | | | | <u>I</u> | | | | | | |
| Myeloma markers<br>(labs)w | | Х | | Х | | | | | | | | | | | Х | | | | Bwks u | | · | oofter until | X |
| | | | | | | | | | | | | | | | | | Qow | ks uni | JI VVK <i>I</i> | ۷, ۷۱ | ZWKS trief | eafter until | PD |
| Bone marrow sample <sup>y, z</sup> | | Xx | | Х | | | | | | | | | | | | | | | Х | Х | Х | | Х |
| Bone survey <sup>aa</sup> | | | | Х | | | | | | | | | | | | | | | | Х | Х | | |
| Research assess | ments | ı | | | 1 | 1 | 1 | 1 | 1 | 1 | | | 1 | 1 | ı | 1 | 1 | | 1 | ı | L | 1 | |
| Pharmaco-<br>genetic - Whole<br>Blood Sample | | | | Xab | | | | | | | | | | | | | | | | | | | |

208470

| | Screening <sup>a</sup> Treatment Phase | | | | | | | | | | | | | | | | DC of | Comple- | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Phase<br>/<br>Eligib<br>Phase | ility | Leukapheresis | Baseline ≤7 days prior to chemo | | | deple<br>erapy | | | T-cell<br>infu-<br>sion | | | | | | | | | | | | Pem-<br>broli-<br>zumab<br>Tx <sup>c</sup> | tion of<br>Treatment<br>Phase or<br>WDd |
| Study Day | Scrn | Elig | | D -14 to<br>D -8 | D -<br>8 | D-7 | D -<br>6 | D -<br>5 | D -<br>4 | D 1 | D2 | D3 | D4 | D5 | Wk<br>1 | Wk<br>2 | W <br>3 | Wk<br>4 | Wk<br>6 | Wk<br>15 | Wk 24<br>&<br>Q12wks | | |
| Window | | | | | | | | | | | | | | | ±1D | ±1D | ±1 | D ±3D | ±3D | ±3D | ±7D | | |
| Bone marrow<br>(bone marrow<br>mononuclear<br>cells) <sup>ac</sup> | | | | X | | | | | | | | | | | | | | | Х | Х | X | | X |
| Cell pheno-typing & Functional assays - PBMC | | | | Х | | | | | | | | | | Х | Х | Х | Х | X | Х | Х | Х | Х | X |
| Vector Copies<br>(Persistence for<br>Research) | | | | Х | | | | | | | | | | Х | Х | Х | Х | X | Х | | | | X |
| Cytokine<br>analyses & Anti-<br>TCR antibodiesp | | | | Х | | | | | | Хр | | Х | | Х | Х | Х | Х | X | Хр | Х | Xp | Х | X |
| cfDNA and exosomes | | Х | | Х | | | | | | | | | | | | | | | Х | Х | Х | | X |

BM = bone marrow; CBC = complete blood count; CMV = cytomegalovirus; CRP = C-reactive protein; DC = discontinuation; DNA = deoxyribonucleic acid; ECHO = echocardiogram; ECOG = Eastern Cooperative Oncology Group; Elig = Eligibility; G-CSF = granulocyte-colony stimulating factor; HBV = hepatitis B virus; HCV = hepatitis C virus; HLA = human leukocyte antigen; HTLV = human T-lymphotropic virus; IMWG = International Myeloma Working Group; MRI = magnetic resonance imaging; MUGA = multiple-gated acquisition scan; PBMC = peripheral blood mononuclear cell; PET = positron emission tomography; PS = Performance Status; RCL = replication competent lentivirus; Scrn = Screening; Tx = treatment; VSV-G = vesicular stomatitis virus envelope glycoprotein; WD = study withdrawal.

a. Written participant informed consent (and participant assent as applicable) must be obtained prior to performing any protocol procedures. An initial Screening informed consent will have been signed prior to obtaining a blood sample for HLA-testing and bone marrow aspirate for antigen testing. The Treatment informed

208470

consent will be signed prior to all other screening procedures. Note: Information regarding ECHO/MUGA scans, and bone surveys which were performed as standard of care assessments within 4 weeks prior to study consent will be acceptable. Laboratory test performed as standard of care and prior to study consent but within 10 days for leukapheresis will be accepted.

- b. Lymphodepleting chemotherapy may only be initiated after the manufactured NY-ESO-1<sup>c259</sup>T-cell product has been received at the site and the bag(s) have passed inspection by site personnel (see further details in study procedures manual [SPM]).
- c. Only for participants enrolled on Arm 2: if participant discontinues from pembrolizumab treatment prior to relapse/progression, this treatment discontinuation visit must be performed including all indicated procedures and assessments listed, unless already recently performed within 30 days. Participant will be maintained in the interventional protocol until disease progression, following the same schedule for safety and disease assessment as Arm 1, and will be transferred to the LTFU protocol ADP-0000-002 as soon as they meet conditions defined under Protocol Section 4.4..
- d. If participant withdraws from the treatment phase prior to disease progression, a completion/withdrawal visit must be performed including all procedures and assessments listed indicated, unless already recently performed within 30 days. All participants will be transferred to the LTFU protocol ADP-0000-002 upon completion/withdrawal from treatment phase as soon as they meet conditions defined under Protocol Section 4.4.
- e. Baseline characteristics include recording time from initial diagnosis and time from last therapy.
- f. Includes prior lines of therapy.
- g. Physical Exam (PE) will only be collected at screening and baseline and every 6 months any abnormal findings outside these time points will be reported as an AE.
- h. Includes concomitant medication since last visit.
- i. Vital signs (temperature, pulse, respirations and blood pressure) on the day of T-cell infusion should be taken pre-infusion; and at 5, 15 and 30 minutes, and 1, 1.5,
- 2, and 4 hours after infusion has started.
- j. Cardiac stress test is performed for participants who are 55 years of age or over (specificity of the test will be at Investigator's discretion).
- k. MUGA and/or ECHO are required at screening. May also be performed post-lymphodepleting chemotherapy if clinically indicated at the discretion of the Investigator.
- 1. Additional tests may be performed at any time if clinically indicated.
- m. Pregnancy test for Female Participant of Reproductive Potential (FSRP) only.
- n. Testing for infectious disease markers is required only at screening and does not need to be repeated at Baseline to satisfy the inclusion / exclusion criteria. Participants who are hepatitis B surface antigen negative but are hepatitis B core antibody positive must have undetectable hepatitis B DNA. Participants who are HCV antibody positive will be screened for HCV RNA by any RT-PCR or bDNA assay.
- o. CMV seropositive participants will continue to be monitored at least every 3 weeks for CMV viremia by CMV DNA PCR until 9 weeks post T-cell infusion (Protocol Section 8.2.3)
- p. Sample for Cytokine levels at Day 1 will be collected pre-infusion. If cytokine release syndrome (CRS) is suspected, cytokine levels as well C-reactive protein levels should be measured approximately every other day until symptoms are improving or an alternative diagnosis is confirmed. Anti-TCR antibodies will be assessed from the same collection as for Cytokines but only at Baseline, Week 6 and Week 24.
- q. Only for participants  $\geq$ 65 years of age.
- r. Refer to Protocol Section 9.1 for instructions and details of AE collection and periods.

- s. Vector Copies (Persistence) and VSV-G DNA (RCL) are Central Labs. Vector copies for safety samples are collected Day1 (pre-infusion) and at Week 15, Week 24, and Week 48 post T-cell infusion, then every 6 months post T-cell infusion from year 2-5, and annually from year 6-15. RCL samples are collected Day1 (pre-infusion), and at Week 15, Week 24, and Week 48 post T-cell infusion, and then annually.
- t. Testing of participant leukapheresis will meet regional legislative requirements. In the EU this may include screening for Treponema pallidum (syphilis), details will be defined in the SPM.
- u. G-CSF will be given from 24 hours after the last dose of cyclophosphamide until resolution of neutropenia in accordance with American Society of Clinical Oncology (ASCO) guidelines or institutional practice. Long-acting (pegylated) G-CSF may be substituted according to institutional practice as described in Protocol Section 8.8.1.
- v. Participants in Arm 2 will receive 200 mg pembrolizumab IV for the first time on Week 3 Subsequent doses will be administered every 3 weeks thereafter up to Week 108. Schedule adjustments are outlined in the protocol (Protocol Section 5.4.1).
- w. SPEP + immunofixation; quantitative IgG, IgM, IgA; UPEP + immunofixation based on 24 hour urine collection; serum free  $\kappa$  and  $\lambda$  light chain levels and  $\kappa/\lambda$  ratio determination; beta-2-microgobulin.
- x. The BM sample is optional for eligibility if participant had prior histological confirmation of the disease.
- y. Bone marrow (BM) sampling should be preferably an aspirate over a fresh biopsy; aspirates are required at Screening, Baseline, as well as for MRD analysis.
- z. BM samples will be obtained at baseline, at Week 15 and at Disease Progression (before starting a new treatment) per standard of care and at the time of a complete response assessment (per IMWG response criteria, see Protocol Section 16.4). If the participant received systemic anticancer therapy between leukapheresis and lymphodepleting chemotherapy for disease control, then the timing of the BM sample at baseline is critical and must respect the wash-out periods of Exclusion criterion #3 (Protocol Section 4.2). A BM sample will also be collected at Week 6. A BM sampling at Week 24 is strongly recommended but not mandatory (per PI's discretion). A BM sampling should also be analyzed at the time of a complete response (CR) assessment as per IMWG criteria (see Protocol Section 16.4), in order to confirm CR. Additional BM samples for research purposes semi-annually (optional) or whenever follow-up marrow collection may be performed at PI's discretion. The BM sample obtained at the time point believed to be the closest to maximum response will be analyzed for Minimal Residual Disease (MRD). Refer to Protocol Section 7.5.3 for further specific details.
- aa. MRI and PET scan if clinically indicated.
- ab. If pharmacogenetics sample collection is not done at baseline, it may be done at any other subsequent visit while the participant is in the treatment phase of the study. Collection of pharmacogenetics sample is optional and all participants who participate must provide consent for pharmacogenetics blood sample collection. ac. Will be conducted every time a BM sample is obtained. Research includes tumor antigen, gene marked T-cells, T-cell clones and cytokines. Cytogenetics should be performed at least at baseline and at relapse.

208470

# 14.2.2. Schedule of Procedures in Long-Term Follow-up prior to Transfer to LTFU Protocol

| Time post-infusion | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Year 1 | | Ye | ar 2 | Ye | ear 3 | Ye | ear 4 | Ye | ear 5 | Years 6-15 |
| Months | 3 | 6 | 12 | 18 | 24 | 30 | 36 | 42 | 48 | 54 | 60 | Annually |
| Visit window | ± 2 w | veeks | ± 3 1 | nonths | | | | | | | | ± 6 months |
| Safety Assessments | | | | | | | | | | | | |
| Medical History and Physical Exam <sup>1</sup> | | X | X | X | X | X | X | X | X | X | X | X |
| Mutagenic agents, other investigational agents or anti-<br>cancer therapies <sup>1</sup> | | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events <sup>2</sup> | | X | X | X | X | X | X | X | X | X | X | X |
| Hematology | | X | X | | X | | X | | X | | X | $X^3$ |
| Serum chemistry | | X | X | | X | | X | | X | | X | $X^3$ |
| Central Lab | | | | | | | | | | | | |
| VSV-G DNA (RCL) for safety <sup>4</sup> | X | X | X | | X | | X | | X | | X | X |
| Vector Copies (Persistence) for safety <sup>5</sup> | X | X | X | X | X | X | X | X | X | X | X | $X^3$ |
| Other Assessments | | | | | | | | | | | | |
| Overall Survival | | X | X | X | X | X | X | X | X | X | X | X |

- 1. New medical history/medications/chemotherapies
- 2. Adverse event collection is limited to:
  - New malignancies
  - New incidence or exacerbation of a pre-existing neurologic disorder
  - New incidence or exacerbation of a prior rheumatologic or other autoimmune disorder
  - New incidence of a hematologic disorder
  - Opportunistic and or serious infections
  - Unanticipated illness and/or hospitalization deemed related to gene modified cell therapy
- 3. In year 6-15, laboratory assessments are performed for as long as persistence is analyzed. If persistence samples are discontinued (Protocol Section 10.3.1 and Section 10.3.2) then laboratory assessments are discontinued.
- 4. Samples for RCL (VSV-G copies) are collected as described in Protocol Section 10.1.1.
- 5. Samples for persistence are collected as described in Protocol Section 10.1.3.1 and Section 10.1.3.2

208470

# 14.3. Appendix 3: Assessment Windows

# 14.3.1. Definitions of Assessment Windows for Analyses

No assessment windows will be applied.

208470

# 14.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 14.4.1. Study Phase

### 14.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | End date of medication is not missing and is before the start date of lymphodepletion OR lymphodepletion chemotherapy start date is missing |
| Concomitant | Any medication that is not a prior |

### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 14.4.1.2. Study Phases for Anti-Cancer Therapy/Surgery

| Study Phase | Definition |
|---|---|
| On-Study | Start date is on or after the first day of lymphodepletion chemotherapy (both start date and lymphodepletion chemotherapy start date not missing). |
| Prior | Not classified as On-Study. |

### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for anti-cancer therapy

The prior phase will be further subdivided as follows:

| Study Phase | Definition |
|---|---|
| Prior to leukapheresis | If classified as prior and entered on the screening visit 2 eCRF |
| Leukapheresis to lymphodepletion | If classified as prior and not entered on the screening visit 2 eCRF. |

#### NOTES:

• Please refer to Appendix 7 for handling of missing and partial dates for anti-cancer therapy

# 14.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date is on or after lymphodepletion chemotherapy start date. (Lymphodepletion Start Date ≤ AE Start Date)</li> <li>If AE onset date is missing and AE end date is before the lymphodepletion start date, then the AE will not be classified as Treatment-Emergent. If AE onset date is missing and AE end date is either missing or on or after lymphodepletion start date, then the AE will be classified as treatment-emergent</li> <li>Partially missing AE onset and end dates will be imputed following rules in Section 14.7.2.1 for determining Treatment Emergent AEs</li> </ul> |

208470

# 14.5. Appendix 5: Data Display Standards & Handling Conventions

# 14.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server : US1SALX00259 | |
| HARP Compound | : arprod\GSK3377794\mid208470 |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.1).</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for SAC. | |

# 14.5.2. Reporting Standards

### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All
  participant level listings should be located in the modular appendices as ICH or non-ICH listings
- While text within this RAP uses the term "participant", all data displays (Tables, Figures, and Listings) will use the term "subject", reflecting CDISC and GSK Data Display Standards terminology.

### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

208470

| Unscheduled Visits | |
|---|---|
| <ul> <li>Unscheduled visits will not be included in summary tables and/or figures, except in cases where<br/>worse-case post-baseline is calculation.</li> </ul> | |
| <ul> <li>All unschedule</li> </ul> | All unscheduled visits will be included in listings. |
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 14.5.3. Reporting Standards for Pharmacokinetic Data

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | All PK parameters will be derived by the PK programmer. No WNL file will be produced. |
| ADPC data file | Persistence data will be captured in ADBIOMRK, and derived persistence parameters will be captured as additional PARAMCD values in ADBIOMRK. No ADPC data file will be created. |
| Descriptive Summary<br>Statistics, Graphical | Example shells for persistence are provided in Appendix 13. |
| Displays and Listings | Refer to IDSL Statistical Principle 6.06.1. |
| | <b>Note:</b> Concentration values will be imputed as per rules in the RAP. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameters to be<br>Derived by PK<br>Programmer | The following PK parameters will be derived by the PK Programmer: Cmax, Tmax, and $AUC_{(0\text{-}28)}$ . |
| Pharmacokinetic Para | Pharmacokinetic Parameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | No. |

208470

# 14.6. Appendix 6: Derived and Transformed Data

### 14.6.1. General

### Multiple Measurements at One Analysis Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- For character variables, if multiple assessments on different days are reported for the same scheduled assessment, then the worst-case assessment for that scheduled assessment will be analysed.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### Study Day

- Calculated as the number of days from T-cell infusion date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < T-cell infusion Date → Study Day = Ref Date T-cell infusion Date
- Ref Date ≥ T-cell infusion Date → Study Day = (Ref Date T-cell infusion Date) + 1

### **Change from Baseline**

- Change from Baseline = Post-Baseline Visit Value Baseline
- % Change from Baseline = 100 x (Post-Baseline Visit Value Baseline) / Baseline
- Maximum Increase/Decrease from Baseline = maximum (Increase/Decrease from Baseline)
- If either the Baseline or Post-Baseline Visit Value is missing, then both Change from Baseline and % Change from Baseline are set to missing

### **Date of New on Study Anti-Cancer Therapy**

- Derived as the earliest date of new systemic anti-cancer therapy
- Missing or partial dates will be imputed for derivation of new anti-cancer therapy following rules specified in Section 14.7.2.1.

# 14.6.2. Study Population

### Age

 For participants with a T-cell infusion date, age is derived using T-cell infusion date as the reference date. For ITT participants without a T-cell Infusion date, date of eligibility for apheresis is used as the reference date.

### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

# Time since Initial Diagnosis to Screening ICF signed

- Time (in months) since initial diagnosis to screening will be calculated below:
- Months since initial diagnosis = (Date of Screening Visit (Screening ICF Signed) Date of Initial diagnosis +1) / 30.4375

208470

### **On-study Treatment Follow-up Time**

- Time (in months) from T-cell infusion to end of follow-up will be calculated below:
- Months of on-study treatment follow-up = (Date of Death/Last Contact T-cell Infusion Date+1) / 30.4375

### **Extent of Exposure (Pembrolizumab)**

Number of days of exposure to Pembrolizumab will be calculated based on the formula:

**Duration on study treatment** is calculated as the minimum of:

- Last treatment stop date first treatment start date + 21
- Date of death first treatment start date + 1
- Participants who did not report a Pembrolizumab start date will be categorised as having zero days of exposure.
- The cumulative actual dose in mg for Pembrolizumab will be based on the formula:

### Cumulative Dose (mg) = Sum of (200 mg \* % of bag infused at each visit)

 Dose intensity (mg/per 3 weeks) for Pembrolizumab is the cumulative actual dose divided by expected duration of exposure in 3 weeks (expected = (last infusion date – first infusion date + 21)/21)

## 14.6.3. Safety

### **Adverse Events**

### Adverse Events of Special Interest (AESIs)

The events of special interest included from protocol Section 9.13 (Adverse Events of Special Interest). This section includes the following events:

- Guillain-Barre Syndrome
- Recurrent Pancytopenia/Aplastic Anaemia
- Immune Effector-Cell Associated Neurotoxicity Syndrome (ICANS)
- Graft versus Host Disease (GVHD)
- Cytokine Release Syndrome (CRS)

### **Duration of AE**

- Calculated as the number of days from AE Start Date to AE Stop Date:
  - AE Start Date = Missing → Elapse Time = Missing
  - AE Stop Date = Missing → Elapse Time = Missing

Otherwise → Elapsed Time = AE Stop Date – AE Start Date + 1

Imputed dates will not be used to calculate AE duration.

### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the following rules will be applied to impute numeric values:
  - If the reported value is "NOT DETECTED" (or some other indicator of such), then impute to 0 (zero).
  - If the reported value is "OLIGOCLONAL POP" (or some other indicator of such), then no
    imputation of a numeric value will be applied.
  - If the reported value is "TRACE" (or some other indicator of such), then no imputation of a numeric value will be applied.

208470

# 14.6.4. **Efficacy**

Refer to Section 7 for endpoint derivation information.

# Secondary Endpoints

### **Date of Last Contact**

- Last date in all SDTM domains
- If patient died, the last contact date should be death date.
- Dates after date of death will be excluded. Future dates will be excluded.
- SDTM domain SE will be excluded and SDTM variables DM.BRTHDTC, MH.MHSTDTC, SV.SVENDTC, SV.SVSTDTC, DM.RFPENDTC, \_ALL\_.ANALDTC, DV.DVDTC, DV.DVSTDTC, and any other external source data dates as necessary will be excluded
- Partial and missing dates will not be imputed for the purpose of deriving date of last contact

208470

# 14.7. Appendix 7: Reporting Standards for Missing Data

### 14.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>A participant will be considered to have completed the treatment phase (as specified in the protocol) at the earliest point of confirmed progressive disease, 108 weeks following NY-ESO-1<sup>c259</sup>T-cell infusion, or death.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 14.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in participant listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| Responder<br>Analysis | For endpoints which determine the percentage of responders, participants with unknown/not evaluable or missing best overall response will be assumed to be non-responders and will be included in the denominator when calculating the percentages. |

### 14.7.2.1. Handling of Missing and Partial Dates

Imputed partial dates can be used to derive study day, duration, or elapsed time variables, unless otherwise specified. However, imputed dates are not used for deriving the last contact date in the overall survival analysis dataset.

Imputed dates will not be displayed in listings. For listings, use the SDTM character date variables and do not show day and duration based on imputed dates. The imputed dates can be used for sorting the data for listings. In addition, partial dates may be imputed for 'slotting' data to study phases or for specific analysis purposes, as outlined below.

The partial date imputation will follow ADaM conventions. The ADaM approach is to populate the numeric date variables with the imputed date and add a flag variable to the dataset that indicates the level of imputation.

The flag variable can contain the values: blank, 'D', 'M', 'Y'.

blank: indicates that no imputation was done

D='Day': indicates that the day portion of the date is imputed

M='Month': indicates that the month and day portions of the date are imputed

Y='Year': indicates that the entire date (year, month, and day) is imputed

# Example of date variables:

XYZDTC\_ - character date variable

XYZDT - numeric date variable

XYZDTFL - flag variable

Details on imputing partial dates for specific datasets are outlined below.

| Element | Reporting Detail | |
|---|---|---|
| General | Partial dates will be | pe displayed as captured in participant listing displays. |
| Adverse<br>Events | appropriate study | adverse events dataset are used for slotting events to the time periods and for sorting in data listings. E recorded in the eCRF will be imputed using the following |
| | Missing start day | <ul> <li>If lymphodepletion start date is missing (i.e. participant did not start lymphodepletion), then set start date = 1st of month.</li> <li>Else if lymphodepletion start date is not missing: <ul> <li>If month and year of start date = month and year of lymphodepletion start date then</li> <li>If stop date contains a full date and stop date is earlier than lymphodepletion start date then set start date= 1st of month.</li> <li>Else set start date = lymphodepletion start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | Missing start day and month | <ul> <li>If lymphodepletion start date is missing (i.e. participant did not start lymphodepletion), then set start date = January 1st.</li> <li>Else if lymphodepletion start date is not missing: <ul> <li>If year of start date = year of lymphodepletion start date then</li> <li>If stop date contains a full date and stop date is earlier than lymphodepletion start date then set start date = January 1st.</li> <li>Else set start date = lymphodepletion start date.</li> <li>Else set start date = January 1st.</li> </ul> </li> </ul> |
| | Missing stop day Missing stop day and month | Last day of the month will be used. No Imputation |
| | Completely missing start/end date | No imputation |
| Anti-Cancer<br>Therapy<br>(including | applied. | ng start or end dates will remain missing, with no imputation e contains a year only set to January 1st. |

| Element | Reporting Detail | |
|---|---|---|
| stem cell<br>transplant)<br>and<br>Radiotherapy | If partial start date | e contains a month and year set to the 1st of the month. end dates will not be imputed. |
| Concomitant Medications/ Blood Supportive Products | <ul><li>concomitant.</li><li>Completely missi</li><li>Partial start dates</li></ul> | rules will be used for classifying a medication as prior or ng start dates will not be imputed. s for any concomitant medications recorded in the eCRF will be e following convention: If lymphodepletion start date is missing (i.e. participant did not |
| | iviissiiig stait day | <ul> <li>If lymphodepletion start date is missing (i.e. participant did not start lymphodepletion), then set start date = 1st of month.</li> <li>Else if lymphodepletion start date is not missing: <ul> <li>If month and year of start date = month and year of lymphodepletion start date then</li> <li>If stop date contains a full date and stop date is earlier than lymphodepletion start date then set start date= 1st of month.</li> <li>Else set start date = lymphodepletion start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | Missing start day and month | <ul> <li>If lymphodepletion start date is missing (i.e. participant did not start lymphodepletion), then set start date = January 1st.</li> <li>Else if lymphodepletion start date is not missing: <ul> <li>If year of start date = year of lymphodepletion start date then</li> <li>If stop date contains a full date and stop date is earlier than lymphodepletion start date then set start date = January 1st.</li> <li>Else set start date = lymphodepletion start date.</li> <li>Else set start date = January 1st.</li> </ul> </li> </ul> |
| | Missing end day Missing end day and month | A '28/29/30/31' will be used for the day (dependent on the month and year) A '31' will be used for the day and 'Dec' will be used for the month. |
| | Completely missing start/end date | No imputation |
| New Anti-<br>Cancer<br>Therapy/<br>Stem cell<br>transplants<br>for Efficacy<br>Evaluation<br>(e.g.,<br>response<br>rate, time to<br>event) | Completely missi Partial start dates If both month If only day is If the month used for If the month used for If the month used for If the month used for If the month used for Otherwise | ng start dates will remain missing, with no imputation applied; swill be imputed using the following convention: and day are missing, no imputation will be applied; missing: onth of partial date is the same as the month of T-cell infusion, of (date of T-cell infusion date + 1, last day of the month) will be the day; onth of partial date is the same as the month of last disease ment and the last disease assessment is PD, minimum of (last date se assessment + 1, last day of the month) will be used for the day; onditions above are met, the later date will be used for the day; se, a '01' will be used for the day; rtial missing end dates will remain missing, with no imputation |

# 14.8. Appendix 8: Values of Potential Clinical Importance

## 14.8.1. Laboratory Values

Reference ranges for all laboratory parameters collected throughout the study are provided by the laboratory. A laboratory value that is outside the reference range is considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Note: a high abnormal or low abnormal laboratory value is not necessarily of clinical concern. The laboratory reference ranges will be provided on the listings of laboratory data. Clinical laboratory test results outside of the reference range will be flagged in the listings.

To identify laboratory values of potential clinical importance, National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.03) will be used to assign grades to the relevant laboratory parameters. NCI-CTCAE v4.03 can be found at http://ctep.cancer.gov/reporting/ctc.html.

For laboratory data which are not listed in the NCI CTCAE v4.03, a summary of values outside the normal range will be provided.

For lab test values that can be graded, values of grade 1 or above are defined as values of potential clinical concern. For lab test values that cannot be graded, values out of the normal range are defined as values of potential clinical concern. For lab tests reported descriptively as 'Normal', 'Abnormal, not clinically significant', or 'Abnormal, clinically significant' (such as urinalysis), responses of 'Abnormal, clinically significant' will be considered as of potential clinical concern.

### 14.8.2. ECG

The following criteria will be used to flag electrocardiogram (ECG) values that are values of potential clinical importance:

To identify QTc (Bazett's or Fridericia's) values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign grades (see adverse event 'Electrocardiogram QT corrected interval prolonged'). The eCRF collects either QTcB or QTcF. Note that there is a slight inconsistency between CTCAE v4 and ICH E14 (Absolute QTc interval prolongation). It was decided to align with CTCAE for the oncology standard categories.

The following criteria will be used to flag other ECG values that are values of potential clinical importance:

| PCI Flag | Potential Clinical Importance (PCI) Range | Unit |
|----------|-------------------------------------------|------|
| High (H) | Grade 2 or Higher (QTc≥481)<br>or | Msec |
| | QTc increase from baseline of >30msec | |

# 14.8.3. Vital Signs

To identify heart rate values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign categories that align with the grades for 'Sinus bradycardia', 'Sinus tachycardia', 'Supraventricular tachycardia', and 'Ventricular tachycardia'.

The following criteria will be used to flag vital sign values that are values of potential clinical importance:

| Vital Sign Parameter | Potential Clinical Importance (PCI) Range | Unit |
|---|---|---|
| Decrease from baseline<br>Heart Rate | Decrease to <60 | bpm |
| Increase from baseline Heart Rate | Increase to >100 | bpm |

To identify blood pressure values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign categories that align with the grades for 'Hypertension'.

| Vital Sign Parameter | Potential Clinical Importance (PCI) Range | Unit |
|--------------------------|-------------------------------------------|------|
| Increase from baseline | ≥120 to <140 (Grade 1) | mmHg |
| Systolic Blood Pressure | ≥140 to <160 (Grade 2) | |
| | ≥160 (Grade 3) | |
| Increase from baseline | ≥80 to <90 (Grade 1) | mmHg |
| Diastolic Blood Pressure | ≥90 to <100 (Grade 2) | |
| | ≥100 (Grade 3) | |

To identify temperature values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign categories that align with the grades for 'Hypothermia' and 'Fever'.

| Vital Sign Parameter | Potential Clinical Importance (PCI) Range | Unit |
|---|---|---|
| Increase from baseline temperature | Increase to ≥38 | Degrees C |
| Decrease from baseline temperature | Decrease to ≤35 | Degrees C |

To identify respiratory rate of potential clinical importance, NCI-CTCAE v4.03 will be used to assign categories that align with the grades for 'Respiratory'.

| Vital Sign Parameter | Potential Clinical Importance (PCI) Range | Unit |
|---|---|---|
| Increase from baseline | Increase to >30 | Breaths/minute |
| respiratory rate | | |
208470

## 14.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

Not applicable.

208470

# 14.10. Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses

Not applicable.

## 14.11. Appendix 11: Abbreviations & Trademarks

## 14.11.1. Abbreviations

| Abbreviation | Description |
|---|---|
| Abbreviation | Description Applying Data Model |
| | Analysis Data Model |
| AECL | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ALT | Alanine Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| AUC | Area Under the Curve |
| BMMC | Bone Marrow Mononuclear Cells |
| BOR | Best Overall Response |
| CDISC | Clinical Data Interchange Standards Consortium |
| Cmax | Peak Expansion |
| CMV | Cytomegalovirus |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CR | Complete Response |
| CRP | C-reactive Protein |
| CRS | Cytokine Release Syndrome |
| CSR | Clinical Study Report |
| CTCAE | Common Toxicity Criteria for Adverse Events |
| DNA | Deoxyribonucleic Acid |
| DBF | Database Freeze |
| DBR | Database Release |
| DoR | Duration of Response |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Record Form |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FLC | Free Light Chain |
| GBS | Guillain-Barre Syndrome |
| G-CSF | Granulocyte-Colony Stimulating Factor |
| GSK | GlaxoSmithKline |
| GvHD | Graft versus Host Disease |
| HLA | Human Leukocyte Antigen |
| IA | Interim Analysis |
| ICANS | Immune Effector-Cell Associated Neurotoxicity Syndrome |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IMWG | International Myeloma Working Group |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| LFT | |
| LFI | Liver Function Test |

208470

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| LTFU | Long-Term Follow-Up |
| mITT | Modified Intent-To-Treat |
| MR | Minimal Response |
| MRD | Minimal Residual Disease |
| NCI | National Cancer Institute |
| NE | Not Evaluable |
| ORR | Overall Response Rate |
| OS | Overall Survival |
| PCI | Potential Clinical Importance |
| PCR | Polymerase Chain Reaction |
| PD | Progression Disease |
| PFS | Progression-free Survival |
| PP | Predictive Probability |
| PR | Partial Response |
| PT | Preferred Term |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RCL | Replication Competent Lentivirus |
| RRMM | Relapsed Refractory Multiple Myeloma |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| sCR | Stringent Complete Response |
| SD | Stable Disease |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| SRT | Safety Review Team |
| TFL | Tables, Figures & Listings |
| TLT | Treatment Limiting Toxicity |
| Tmax | Time to Peak Expansion |
| TTR | Time to Response |
| ULN | Upper Limit of Normal |
| VGPR | Very Good Partial Response |

## 14.11.2. Trademarks

| Tra | ademarks of the GlaxoSmithKline<br>Group of Companies |
|-----|-------------------------------------------------------|
| KEY | TRUDA |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| SAS |
| WinNonlin |

208470

#### 14.12. Appendix 12: List of Data Displays

#### 14.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|------------------|------------------|
| Study Population | 1.0010 to 1.0220 | NA |
| Efficacy | 2.0010 to 2.0020 | 2.0030 to 2.0070 |
| Safety | 3.0010 to 3.0620 | 3.0630 to 3.0680 |
| Biomarker | 3.0690 to 3.0690 | NA |
| Pharmacokinetic | 4.0010 to 4.0020 | 4.0030 to 4.0050 |
| Section | Listir | ngs |
| ICH Listings | 0010 to | 0430 |
| Other Listings | 0440 to 0520 | |

### 14.12.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 13: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Biomarker | BIO_Fn | BIO_Tn | BIO_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

#### 14.12.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

208470

# 14.12.4. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subject | Disposition | | | | |
| 1.0010 | mITT | [Non-Standard]<br>POP_T2 | Summary of Subject Status – Treatment Phase (mITT) | ICH E3, FDAAA, EudraCT Subject Status: Completed, Ongoing, Did not complete. Use reasons on the EOT CRF (reason for early discontinuation) for withdrawal, prepopulate all of them in the display. Note that progressive disease, death, and not progressed at 108 weeks are the only reasons for completion of the treatment phase. Not aligned w/study 208469 (MRCLS). | SAC |
| 1.0020 | mITT | [Non-Standard]<br>POP_T3 | Summary of Subject Status – End of Study (mITT) | ICH E3, FDAAA, EudraCT Use logic provided in RAP text to derive end-of-study status. Subject Status: Completed, Ongoing, Withdrawn Reason for withdrawal comes from treatment phase table above. Not aligned w/study 208469 (MRCLS). | SAC |
| 1.0030 | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements Align w/study 208469 (MRCLS). | SAC |
| 1.0040 | ITT | SD4 | Summary of Reasons for Study Treatment Discontinuation (Pembrolizumab) | Only include participants from Arm 2. Reasons for discontinuation should match the Pembrolizumab disposition eCRF in content and order Not aligned w/ 208469 (MRCLS) | SAC |

| Study P | opulation Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.0050 | Enrolled | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations<br>Align w/study 208469 (MRCLS). | SAC |
| Populat | ion Analysed | | | | |
| 1.0060 | Screened | SP1A | Summary of Study Populations | IDSL<br>Screened, Enrolled, ITT, mITT only.<br>Align w/study 208469 (MRCLS). | SAC |
| Protoco | l Deviations | | | | |
| 1.0070 | ITT | DV1 | Summary of Important Protocol Deviations | ICH E3<br>Align w/study 208469 (MRCLS). | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.0080 | mITT | DM1 | Summary of Demographic Characteristics (mITT) | ICH E3, FDAAA, EudraCT Report baseline height, weight, BMI, and BSA. Report Race but not Race Detail. Age groups to be presented: <=18, 19-64, and >=65 years. Align w/study 208469 (MRCLS). | SAC |
| 1.0090 | Enrolled | DM11 | Summary of Age Ranges | EudraCT Age groups to be presented: 18-64, 65-84 and >=85 years. Align w/study 208469 (MRCLS). | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Disease | <b>Characteristic</b> | cs | | | |
| 1.0100 | mITT | DC1 | Summary of Disease Characteristics at Initial Diagnosis (mITT) | ICH E3 Time from initial diagnosis to screening ICF signed (in months), stage at diagnosis, histologic type, % clonal bone marrow plasma cells, presence and type of end organ damage, presence and type of plasmacytoma, and chromosomal aberrations (previously referred to as karyotype). Not aligned w/study 208469 (MRCLS). | SAC |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.0110 | mITT | DC2 | Summary of Disease Characteristics at Screening (mITT) | ICH E3 Type of multiple myeloma (IgA Kappa, IgA Lambda, IgG Kappa, etc.), HLA status (Allele 1 & Allele 2), NY-ESO-1 status, LAGE-1a status, number of radiotherapy regimens prior to leukapheresis, number of systemic therapy regimens prior to leukapheresis, receipt of stem-cell transplant prior to leukapheresis (Y/N), bone lesion (Y/N), and subtype of stem-cell transplant received (autologous or allogeneic). Break down "Number of Prior Systemic Therapy Regimens" into {0,1,2,3,4,5,6,>6}. Also, use the new derivation of lines of systemic therapy (i.e., count systemic therapy + conditioning chemo associated w/stem cell therapy) – please add a footnote that makes this clear. Not aligned w/study 208469 (MRCLS). | SAC |
| Medical | Medical Conditions and Concomitant Medications | | | | |
| 1.0120 | mITT | MH4 | Summary of Medical Conditions (mITT) | ICH E3 Include both past and ongoing medical conditions at screening. Align w/study 208469 (MRCLS). | SAC |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.0130 | mITT | CM8 | Summary of Concomitant Medications (mITT) | ICH E3 Use GSK Drug Coding Dictionary Align w/study 208469 (MRCLS). | SAC |
| 1.0140 | mITT | BP1A | Summary of Blood Products on Treatment (mITT) | Using the same rule as con meds, include only "concomitant blood products" in the display and provide a footnote that explains this clearly. Align w/study 208469 (MRCLS). | SAC |
| Anti-Ca | ncer Therapy | | | | |
| 1.0150 | mITT | AC1 | Summary of Prior Anti-Cancer Therapy (mITT) | IDSL In addition to prior systemic and radiation therapies, please include prior stem cell therapy (by subtype: autologous or allogeneic) in this summary. Systemic therapy should include prior to leukapheresis + full line of therapy starting after leukapheresis, and radiotherapy and surgery should include prior to lymphodepletion. Add footnote: "Note: Includes all anticancer therapy prior to lymphodepletion except bridging therapies." With the exception of stem cell being included, this display should align w/study 208469 (MRCLS). | SAC |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.0160 | mITT | FAC1 | Summary of On-Study Anti-Cancer Therapy (mITT) | IDSL Add time from T-cell infusion to the first post-treatment anti-cancer therapy. In addition to systemic and radiation therapies, please include stem cell therapy (by subtype: autologous or allogeneic) in this summary. With the exception of stem cell being included, this display should align w/study 208469 (MRCLS). | SAC |
| 1.0170 | mITT | CM1 | Summary of Prior Dictionary Coded Anti-Cancer Therapy (mITT) | IDSL Use GSK Drug Coding Dictionary Systemic therapy should include prior to leukapheresis + full line of therapy starting after leukapheresis, and radiotherapy should include prior to lymphodepletion. Note that while stem cell therapy is not included in this summary, conditioning chemotherapy for the stem cell therapy is included. Add footnote: "Note: Includes all anti- cancer therapy prior to lymphodepletion except bridging therapies." Add footnote: "Note: Stem cell therapy is not included in this summary." Align w/study 208469 (MRCLS). | SAC |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.0180 | mITT | AC3 | Summary of Number of Prior Anti-Cancer Therapy Regimens (mITT) | IDSL Summarize all prior systemic therapy and radiotherapy regimens prior to lymphodepletion. Do not split out by type of systemic regimen as multiple types could make up a regimen. Add footnote: "Note: Includes all anticancer therapy prior to lymphodepletion except bridging therapies." Not aligned w/study 208469 (MRCLS) | SAC |
| 1.0190 | mITT | CM1 | Summary of On-Study Dictionary Coded Anti-Cancer Therapy (mITT) | IDSL Use GSK Drug Coding Dictionary Note that while stem cell therapy is not included in this summary, conditioning chemotherapy for the stem cell therapy should be included. Add footnote: "Note: Stem cell therapy is not included in this summary." Align w/study 208469 (MRCLS). | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.0200 | mITT | CM1 | Summary of Bridging Therapy (mITT) | IDSL Summarize all prior therapies identified as bridging. In addition to systemic and radiation therapies, please include prior stem cell therapy in this summary. With the exception of stem cell being included, this display should align w/study 208469 (MRCLS). Add footnote: "Note: Includes all anticancer therapy initiated between leukapheresis and lymphodepletion identified as bridging." | SAC |
| Exposu | ıre | | | | |
| 1.0210 | mITT | OEX1 | Summary of Total Infused Transduced T-cells | Report total number of infused transduced T-cells in 10^9 cells and categorize it into: <1, >=1 to <=8, >8 and <1, >=1 to <=3, >3 to <=8, >8 Align w/study 208469 (MRCLS). | SAC |
| 1.0220 | mITT | [Non-Standard]<br>POP_T1 | Summary of Leukapheresis, Lymphodepletion, T-cell Infusion, and Pembrolizumab Administration | Add number of subjects infused with minimum dose of 1 x 10^9 transduced cells (i.e., in addition to the total number who underwent infusion). Please add a line for Pembro. Not aligned w/study 208469 (MRCLS). | SAC |

208470

# 14.12.5. Efficacy Tables

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Overall | Response Rat | e (ORR) | | | |
| 2.0010 | mITT | RE1a | Summary of Investigator-Assessed Best Response with Confirmation (IMWG 2016) (mITT) | Add Total column. Add Overall Response (sCR + CR + VGPR + PR) and include 95% CI for Overall Response Rate. Omit all hypothesis testing sections. Not aligned w/study 208469 (MRCLS). | SAC |
| Time to | Event | | | | |
| 2.0020 | mITT | TTE1 | Summary of Investigator-Assessed Progression Free Survival (IMWG 2016) | Unit = months. Include a Total column. Only create if at least 3 subjects in the study Omit all hypothesis testing sections i.e., Hazard Ratio estimate and 95%CI (marked as optional in IDSL shell). Include footnote: "Note: Progression Free Survival is defined as the interval between the date of T-cell infusion and the date of confirmed progressive disease or death per IMWG 2016." Align w/study 208469 (MRCLS). | SAC |

#### 208470

# 14.12.6. Efficacy Figures

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Respor | ses by Myelor | na Biomarkers | | | |
| 2.0030 | mITT | [Non-Standard]<br>EFF_F1 | Percent Change at Maximum Reduction from Baseline in M-Protein or Serum Free Light Chain (FLC) Measurement | Waterfall plot. Use Serum M-protein, Urine-M-protein (if no Serum M-protein) and difference between 2 types of Serum FLC (if Serum M-protein and Urine M-protein not available), as relevant per subject. Do not report separately by arm; rather, include all subjects on the same plot. Color the bars by "Type of Myeloma Marker" and "Treatment Arm". Example: Arm 1 Serum M prot='Solid Blue', Arm 2 Serum M prot='Striped Blue'. Not aligned w/study 208469 (MRCLS). | SAC |
| 2.0040 | mlTT | [Non-Standard]<br>EFF_F2 | Spider Plot of Percent Change from Baseline in Myeloma<br>Biomarkers by Subject | Create a separate plot for each subject, showing on each plot: Serum M-protein, Urine-M-protein and difference between 2 types of Serum FLC. Include date of first pembro dose on the plot for each subject. Not aligned w/study 208469 (MRCLS). | SAC |
| 2.0050 | mITT | [Non-Standard]<br>EFF_F2 | Composite Spider Plot of Percent Change from Baseline in Myeloma Biomarkers for All Subjects | Create a composite plot, with all subjects included (1 line per subject). The line for each subject will represent the subject's "chosen marker" from the waterfall plot above. Include date of first pembro dose on the plot for each subject. | SAC |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Not aligned w/study 208469 (MRCLS). | |
| Time to | Event | | | | |
| 2.0060 | mITT | TTE10 | Graph of Kaplan-Meier Curve of Investigator-Assessed Progression Free Survival with 95% Confidence Band by Treatment Arm (IMWG 2016) | Unit = months. Create separate KM curves (lines) for treatment arms (distinguish lines by color or pattern). Only create if at least 3 subjects in a single arm. Similar to the footnote used in DoR displays, add a footnote that defines PFS as including confirmed progressive disease. Align w/study 208469 (MRCLS). | SAC |
| 2.0070 | mITT | TTE10 | Graph of Kaplan-Meier Curve of Investigator-Assessed Progression Free Survival with 95% Confidence Band for All Subjects (IMWG 2016) | Unit = months. Create single KM curve for all subjects. Only create if at least 3 subjects overall in the study. Similar to the footnote used in DoR displays, add a footnote that defines PFS as including confirmed progressive disease. Align w/study 208469 (MRCLS). | SAC |

#### 208470

# 14.12.7. Safety Tables

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Adverse I | Events (AEs) | | | | |
| 3.0010 | ITT | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 Add Total column. Do not use combined PTs. Align w/study 208469 (MRCLS). | SAC |
| 3.0020 | mITT | AE1 | Summary of All Treatment Emergent Adverse Events by System Organ Class and Preferred Term | ICH E3 Add Total column. Do not use combined PTs. Treatment emergent only. Align w/study 208469 (MRCLS). | SAC |
| 3.0030 | ITT | OAE07 | Summary of All Adverse Events by Maximum Grade<br>Separately for Treatment Arms and Overall | Add total "by group" page (i.e., subheading should be "Treatment: Total (N=XXX)"). Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as column header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. Align w/study 208469 (MRCLS). | SAC |
| 3.0040 | ITT | AE18 | Summary of All Adverse Events by Maximum Grade and Treatment Arm | Include Total column. Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as column header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. | SAC |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.0050 | mITT | OAE07 | Summary of All Treatment Emergent Adverse Events by Maximum Grade Separately for Treatment Arms and Overall | Treatment emergent only. Add total "by group" page (i.e., subheading should be "Treatment: Total (N=XXX)"). Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as column header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. Align w/study 208469 (MRCLS). | SAC |
| 3.0060 | mITT | AE18 | Summary of All Treatment Emergent Adverse Events by Maximum Grade and Treatment Arm | Treatment emergent only. Include Total column. Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as column header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. | SAC |
| 3.0070 | mITT | OAE07 | Summary of All Study-Treatment Related Adverse Events by Maximum Grade Separately for Treatment Arms and Overall | ICH E3 Treatment emergent only. Add total by-group page. Treatment related, including lymphodepleting chemotherapy, T-cell infusion, and pembrolizumab. Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as column header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. Align w/study 208469 (MRCLS). | SAC |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.0080 | mITT | AE18 | Summary of All Study-Treatment Related Adverse Events by Maximum Grade and Treatment Arm | ICH E3 Treatment emergent only. Include Total column. Treatment related, including lymphodepleting chemotherapy, T-cell infusion, and pembrolizumab. Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as column header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. | SAC |
| 3.0090 | mITT | OAE07 | Summary of All T-Cell Infusion Related Adverse Events by Maximum Grade Separately for Treatment Arm and Overall | ICH E3 Treatment emergent only. Add total by-group page. Treatment related (T-cell infusion). Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as column header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. Align w/study 208469 (MRCLS). | SAC |
| 3.0100 | mITT | AE18 | Summary of All T-Cell Infusion Related Adverse Events by Maximum Grade and Treatment Arm | ICH E3 Treatment emergent only. Include Total column. Treatment related (T-cell infusion). Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as column header. | SAC |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Present grades 3+4+5 combined (as in OAE01) rather than 3+4. | |
| 3.0110 | mITT | OAE07 | Summary of All Lymphodepletion-Related Adverse Events by Maximum Grade Separately for Treatment Arm and Overall | ICH E3 Treatment emergent only. Add total by-group page. Treatment related (lymphodepleting chemotherapy). Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as column header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. Align w/study 208469 (MRCLS). | SAC |
| 3.0120 | mITT | AE18 | Summary of All Lymphodepletion-Related Adverse Events by Maximum Grade and Treatment Arm | ICH E3 Treatment emergent only. Include Total column. Treatment related (lymphodepleting chemotherapy). Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as column header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. | SAC |
| 3.0130 | ITT | OAE07 | Summary of All Serious Adverse Events by Maximum Grade Separately for Treatment Arm and Overall | ICH E3 Treatment emergent only. Serious events. Add total by-group page. Use combined PTs with footnote "Preferred terms are combined." | SAC |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Use "Adverse Event" (rather than "Preferred Term") as column header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. Align w/study 208469 (MRCLS). | |
| 3.0140 | ITT | AE18 | Summary of All Serious Adverse Events by Maximum Grade and Treatment Arm | ICH E3 Treatment emergent only. Serious events. Include Total column. Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as column header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. | SAC |
| 3.0150 | ITT | AE15 | Summary of All Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT Add Total column. Do not combine Preferred Terms. Align w/study 208469 (MRCLS). | SAC |
| 3.0160 | ITT | AE3 | Summary of All Non-Serious Study-Treatment Related AEs by Overall Frequency | Add Total column. Do not combine Preferred Terms. Align w/study 208469 (MRCLS). | SAC |
| 3.0170 | ITT | AE1 | Summary of Adverse Events Grouped by Similarity of Preferred Terms | Add Total column. Use combined PTs with footnote "Preferred terms are combined." Remove overall "ANY EVENT" and synonym level "Any Event" rows. SOC from AE1 should be combined PT. PT from AE1 should be the MEDDRA PT. | SAC |

| Safety: Ta | ables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Label column "Synonym/Preferred<br>Term" rather than "System Organ<br>Class/Preferred Term" (where / indicates<br>new line and indent as in AE1). | |
| | | | | If combined AE does not appear then include a 0 count. Align w/study 208469 (MRCLS). | |
| Adverse I | Events of Spec | ial Interest (AE of | SI) | | |
| 3.0180 | mITT | OAE01 | Summary of Treatment Emergent Adverse Events of Special Interest by Maximum Grade (Focused List) | Treatment emergent only. Add total by-group page (i.e., subheading should be "Treatment: Total (N=XXX)"). Use combined PT identified in the focused list with footnote "Preferred terms are combined". Use "Adverse Event" (rather than "Preferred Term") as column header. Replace SOC with AESI category (use AESI category names from current SRT AESI specification document if these differ to those in RAP). Align w/study 208469 (MRCLS). | SAC |
| 3.0190 | mITT | OAE01 | Summary of Treatment Emergent Adverse Events of Special Interest by Maximum Grade (Comprehensive List) | Treatment emergent only. Add total by-group page (i.e., subheading should be "Treatment: Total (N=XXX)"). Do not use combined PTs. | SAC |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Replace SOC with AESI category (use AESI category names from current SRT AESI specification document if these differ to those in RAP). | |
| 3.0200 | mITT | ESI1 | Summary of Characteristics of Haematopoietic Cytopenias (Focused List) | Align w/study 208469 (MRCLS). Treatment emergent only. Add total column. Use Focused Scope List. Footnote – "Preferred terms identified in the Focused list are summarized". Report for all subjects and for all subjects with event. Report characteristics, outcome, number of occurrences and max grade. Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). | SAC |
| 3.0210 | mITT | ESI1 | Summary of Characteristics of Cytokine Release Syndrome (CRS) | Treatment emergent only. Add total column. Use Focused Scope List. Footnote – "Preferred terms identified in the Focused list are summarized". Report for all subjects and for all subjects with event. Report characteristics, outcome, number of occurrences and max grade. Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). | SAC |
| 3.0220 | mITT | ESI2a | Summary of Onset and Duration of the First Occurrence of Haematopoietic Cytopenias (Focused List) | Treatment emergent only. Add total column. Use Focused Scope List. | SAC |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Footnote – "Preferred terms identified in the Focused list are summarized". Time to onset (days) (-81, 1 -14, 15-30, 31-60, >60). Remove subjects at risk. Duration (days) (1-30,31-90, >90). Onset from first T-cell infusion. Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). Important: The AE collapsing rules of MRCLS should be used for all onset/duration tables, where applicable. | |
| 3.0230 | mITT | ESI2a | Summary of Onset and Duration of the First Occurrence of Haematopoietic Cytopenias (Neutropenia) | Treatment emergent only. Add total column. Use Focused Scope Neutropenia List. Footnote – "Preferred terms identified in the Focused neutropenia list are summarized". Time to onset (days) (-81, 1 -14, 15-30, 31-60, >60). Remove subjects at risk. Duration (days) (1-30,31-90, >90). Onset from first T-cell infusion. Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). Important: The AE collapsing rules of MRCLS should be used for all onset/duration tables, where applicable. | SAC |
| 3.0240 | mITT | ESI2a | Summary of Onset and Duration of the First Occurrence of Haematopoietic Cytopenias (Thrombocytopenia) | Treatment emergent only. Add total column. | SAC |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Use Focused Scope Thrombocytopenia List. Footnote – "Preferred terms identified in the Focused Thrombocytopenia list are summarized". Time to onset (days) (-81, 1 -14, 15- 30, 31-60, >60). Remove subjects at risk. Duration (days) (1-30,31-90, >90). Onset from first T-cell infusion. Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). Important: The AE collapsing rules of MRCLS should be used for all onset/duration tables, where applicable. | |
| 3.0250 | mITT | ESI2a | Summary of Onset and Duration of the First Occurrence of Haematopoietic Cytopenias (Anemia) | Treatment emergent only. Add total column. Use Focused Scope Anemia List. Footnote – "Preferred terms identified in the Focused Anemia list are summarized". Time to onset (days) (-81, 1 -14, 15-30, 31-60, >60). Remove subjects at risk. Duration (days) (1-30,31-90, >90). Onset from first T-cell infusion. Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). Important: The AE collapsing rules of MRCLS should be used for all onset/duration tables, where applicable. | SAC |

| Safety: Ta | ables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.0260 | mITT | ESI2a | Summary of Onset and Duration of the First Occurrence of Cytokine Release Syndrome (CRS) | Treatment emergent only. Add total column. Use Focused Scope List. Footnote – "Preferred terms identified in the Focused list are summarized". Time to onset (days) (-81, 1 -14, 15-30, 31-60, >60). Remove subjects at risk. Duration (days) (1-30, 31-90, >90). Onset from first T-cell infusion. Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). Important: The AE collapsing rules of MRCLS should be used for all onset/duration tables, where applicable. | SAC |
| 3.0270 | mITT | ESI2a | Summary of Onset and Duration of the Last Occurrence of Haematopoietic Cytopenias (Focused List) | Treatment emergent only. Add total column. Use Focused Scope List. Footnote – "Preferred terms identified in the Focused list are summarized". Time to onset (days) (-81, 1 -14, 15-30, 31-60, >60). Remove subjects at risk. Duration (days) (1-30 31-90, >90). Onset from first T-cell infusion. Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). | SAC |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Important: The AE collapsing rules of MRCLS should be used for all onset/duration tables, where applicable. | |
| 3.0280 | mITT | [Non-Standard]<br>SAFE_T1 | Summary of Time to Resolution and Recurrence of Grade 3 and Above Haematopoietic Cytopenias (Focused List) | Treatment emergent only. Use Focused Scope List. Footnote – "Preferred terms identified in the Focused list are summarized". Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). | SAC |
| 3.0290 | mITT | [Non-Standard]<br>SAFE_T1 | Summary of Time to Resolution and Recurrence of Grade 3 and Above Haematopoietic Cytopenias (Neutropenia) | Treatment emergent only. Use Comprehensive Scope List. Footnote – "Preferred terms identified in the Neutropenia focused list are summarized". Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). | SAC |
| 3.0300 | mITT | [Non-Standard]<br>SAFE_T1 | Summary of Time to Resolution and Recurrence of Grade 3 and Above Haematopoietic Cytopenias (Thrombocytopenia) | Treatment emergent only. Use Comprehensive Scope List. Footnote – "Preferred terms identified in the thrombocytopenia focused list are summarized". Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). | SAC |
| 3.0310 | mITT | [Non-Standard]<br>SAFE_T1 | Summary of Time to Resolution and Recurrence of Grade 3 and Above Haematopoietic Cytopenias (Anemia) | Treatment emergent only. Use Comprehensive Scope List. Footnote – "Preferred terms identified in the Anemia focused list are summarized". | SAC |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Do not create if 1 or fewer subjects have event (default to listing). Align w/study 208469 (MRCLS). | |
| Serious a | nd Other Signi | ficant Adverse Ev | ents | | |
| 3.0320 | ITT | AE16 | Summary of All Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT Add Total column. Do not use combined PTs. Align w/study 208469 (MRCLS). | SAC |
| 3.0330 | ITT | OAE07 | Summary of All Serious Adverse Events by Maximum Grade | Add total "by group" page. Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. Align w/study 208469 (MRCLS). | SAC |
| 3.0340 | mITT | OAE07 | Summary of All Serious Treatment Emergent Adverse Events by Maximum Grade Separately for Treatment Arm and Overall | Treatment emergent only. Add total "by group" page. Use combined PTs with footnote "Preferred terms are combined." Use "Adverse Event" (rather than "Preferred Term") as header. Present grades 3+4+5 combined (as in OAE01) rather than 3+4. Align w/study 208469 (MRCLS). | SAC |
| 3.0350 | mITT | AE18 | Summary of All Serious Treatment Emergent Adverse Events by Maximum Grade and Treatment Arm | Treatment emergent only. Use combined PTs with footnote "Preferred terms are combined." | SAC |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Use "Adverse Event" (rather than | |
| | | | | "Preferred Term") as header. | |
| | | | | Present grades 3+4+5 combined (as in | |
| | | | | OAE01) rather than 3+4. | |
| | | | | Align w/study 208469 (MRCLS). | |
| | | | | Treatment emergent only. | |
| | | | | Add total "by group" page. | |
| | | | | Use combined PTs with footnote | |
| | | mill $ \cap \triangle \vdash \cap A \vdash A \vdash$ | Summary of All Study-Treatment Related Serious Adverse Events by Maximum Grade | "Preferred terms are combined." | |
| 3.0360 | mITT | | | Use "Adverse Event" (rather than | SAC |
| | | | | "Preferred Term") as header. | |
| | | | | Present grades 3+4+5 combined (as in | |
| | | | | OAE01) rather than 3+4. | |
| | | | | Align w/study 208469 (MRCLS). | |
| | | | | Treatment emergent only. | |
| | | | | Add total "by group" page. | |
| | | | | Use combined PTs with footnote | |
| | | | Summary of All T-cell Infusion Serious Adverse Events by | "Preferred terms are combined." | |
| 3.0370 | mlTT | OAE07 | Maximum Grade | Use "Adverse Event" (rather than | SAC |
| | | | Maximum Grado | "Preferred Term") as header. | |
| | | | | Present grades 3+4+5 combined (as in | |
| | | | | OAE01) rather than 3+4. | |
| | | | | Align w/study 208469 (MRCLS). | |
| | | | | Treatment emergent only. | |
| 3.0380 | mITT | OAE07 | Summary of All Lymphodepletion-Related Serious Adverse Events by Maximum Grade | Add total "by group" page. | SAC |
| 0.0000 | | 0,120, | | Use combined PTs with footnote | |
| | | | | "Preferred terms are combined." | |

| Safety: Ta | ables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Use "Adverse Event" (rather than | |
| | | | | "Preferred Term") as header. | |
| | | | | Present grades 3+4+5 combined (as in | |
| | | | | OAE01) rather than 3+4. | |
| | | | | Align w/study 208469 (MRCLS). | |
| 3.0390 | ITT | AE3 | Summary of Fatal Adverse Events by Preferred Term | Add Total column. Do not produce if <5 subjects have fatal AE. Do not use combined PTs. Align w/study 208469 (MRCLS). | SAC |
| | | | | Treatment emergent only. | |
| | | | | Add Total column. | |
| | | | | Use combined PTs with footnote | |
| 3.0400 | mITT | AE3 | Summary of Study-Treatment Related Fatal Adverse Events | "Preferred terms are combined." | SAC |
| | | | | Use "Adverse Event" (rather than | |
| | | | | "Preferred Term") as header. | |
| | | | | Align w/study 208469 (MRCLS). | |
| 3.0410 | ITT | AE3 | Summary of All Serious Study-Treatment Related AEs by<br>Overall Frequency | Add Total column. Do not use combined PTs. Align w/study 208469 (MRCLS). | SAC |
| Deaths | | | | | |
| | | | | IDSL | |
| | | | | Add Total column. | |
| 3.0420 | mITT | DD1 | Summary of Deaths | Report time from T-cell infusion to death with median, min, max, 1st Q, 3rd Q in months, >30 days or <=30 days. | SAC |
| | | | | Only report Alive at Last Contact (do not report follow up ongoing/ended). | |

| Safety: Ta | ables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Report primary cause of death categories corresponding to those captured on MM Combo eCRF. Align w/study 208469 (MRCLS). | |
| Laborator | ry: Chemistry | | | | |
| 3.0430 | mITT | LB1 | Summary of Chemistry Changes from Baseline | ICH E3. Add total panel. Align w/study 208469 (MRCLS). | SAC |
| 3.0440 | mITT | OLB9C | Summary of Worst-Case Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3 Include total panel. Report Week 4 and Week 15 visits plus Worst-case post-baseline only. For labs that are gradable by CTCAE v4.03. Align w/study 208469 (MRCLS). | SAC |
| 3.0450 | mITT | OLB11C | Summary of Worst-Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 Include total panel. Do not report by visit. For labs that are NOT gradable by CTCAE v4.03. Add footnote "Only tests that are not gradable by CTCAE are summarized." Align w/study 208469 (MRCLS). | SAC |
| Laborator | ry: Hematology | | 1 | 1 0 | |
| 3.0460 | mITT | LB1 | Summary of Hematology Changes from Baseline | ICH E3. Add total panel. Align w/study 208469 (MRCLS). | SAC |

| Safety: Ta | ables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.0470 | mITT | OLB9C | Summary of Worst-Case Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3 Include total panel. Report Week 4 and Week 15 visits plus Worst-case post-baseline only. For labs that are gradable by CTCAE v4.03. Align w/study 208469 (MRCLS). | SAC |
| 3.0480 | mITT | OLB11C | Summary of Worst-Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 Include total panel. Report Week 4 and Week 15 visits plus Worst-case post-baseline only. For labs that are NOT gradable by CTCAE v4.03. Add footnote "Only tests that are not gradable by CTCAE are summarized." Align w/study 208469 (MRCLS). | SAC |
| Laborator | ry: Other Tests | | | | |
| 3.0490 | mITT | LB1 | Summary of Other Laboratory Changes from Baseline | ICH E3 Add total panel. Include all "other" (non-chemistry, non-hematology) quantitative lab tests (i.e., coagulation, immunology, endocrine, urinalysis, and biomarker). Align w/study 208469 (MRCLS). | SAC |
| 3.0500 | mITT | OBL9C | Summary of Worst-Case Other Laboratory Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3 Include total panel. Report Week 4 and Week 15 visits plus Worst-case post-baseline only. For labs that are gradable by CTCAE v4.03. | SAC |

| Safety: Ta | ables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Include all "other" (non-chemistry, non-hematology) quantitative lab tests (i.e., coagulation, immunology, endocrine, urinalysis, and biomarker). Align w/study 208469 (MRCLS). | |
| 3.0510 | mITT | OLB11C | Summary of Worst-Case Other Laboratory Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 Include total panel. Do not report by visit. For labs that are NOT gradable by CTCAE v4.03. Add footnote "Only tests that are not gradable by CTCAE are summarized." Include all "other" (non-chemistry, non-hematology) quantitative lab tests (i.e., coagulation, immunology, endocrine, urinalysis, and biomarker). Align w/study 208469 (MRCLS). | SAC |
| Performa | nce Status | | | | |
| 3.0520 | mITT | PS1A | Summary of ECOG Performance Status | ICH E3 Add Total column. Only summarize baseline and last assessment. Align w/study 208469 (MRCLS). | SAC |
| 3.0530 | mITT | PS3A | Summary of Change in ECOG Performance Status from Baseline | ICH E3 Add Total column. Include best and worst case. Align w/study 208469 (MRCLS). | SAC |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| ECG | | | | | |
| 3.0540 | mITT | EG1 | Summary of ECG Findings | IDSL Add Total column. "Clinically significant change from baseline" in this standard shell is not collected in this study so cannot be reported; drop from the display. Align w/study 208469 (MRCLS). | SAC |
| 3.0550 | mITT | OECG1C | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | IDSL Include total panel. Do not report by visit. QTcB and QTcF should be reported in this same table but summarized separately. QTcB and QTcF values should not be derived. Align w/study 208469 (MRCLS). | SAC |
| 3.0560 | mITT | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL Include total panel. QTcB and QTcF should be reported in this same table but summarized separately. Align w/study 208469 (MRCLS). | SAC |
| 3.0570 | mITT | OECG2C | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | IDSL Include total panel. Do not report by visit. | SAC |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | QTcB and QTcF should be reported in this same table but summarized separately. Align w/study 208469 (MRCLS). | |
| Vital Sign | s | | | | |
| 3.0580 | mITT | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 Include total panel. Include weight, temp, DBP, SBP pulse rate, respiratory rate. Align w/study 208469 (MRCLS). | SAC |
| 3.0590 | mITT | OVT1C | Summary of Worst-Case Heart Rate Results Relative to Normal Range Post-Baseline Relative to Baseline | IDSL Include total panel. Do not summarize by visit. Align w/study 208469 (MRCLS). | SAC |
| 3.0600 | mITT | OVT2C | Summary of Worst-Case Blood Pressure Results by Maximum Grade Increase Post-Baseline Relative to Baseline | IDSL Include total panel. Do not summarize by visit. Align w/study 208469 (MRCLS). | SAC |
| Replication | on Competent L | _entivirus (RCL) | | | |
| 3.0610 | mITT | [Non-Standard]<br>SAFE_T3 | Summary of Replication Competent Lentivirus Positive | Please produce even if positive counts are low or zero. Align w/study 208469 (MRCLS). | SAC |
| 3.0620 | mITT | [Non-Standard]<br>SAFE_T3 | Summary of Subjects Showing >1% Gene Marked PBMCs 1<br>Year Post-Treatment | Define 1 year conservatively as at least 360 days since infusion or month 12 visit. Align w/study 208469 (MRCLS). | SAC |

#### 208470

# 14.12.8. Safety Figures

| Safety: | Safety: Figures | | | | | | | | |
|---|---|---|---|---|---|--|--|--|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable | | | | |
| Duration Plots | | | | | | | | | |
| 3.0630 | mlTT | [Non-Standard]<br>SAFE_F2 | Plot of Duration on Treatment Phase | (1) Show all subjects on the same plot; do not show by treatment arm. Instead, add Arm label as an additional column to the right of Age/Sex. (2) Sort the Subject ID (y-axis) in ascending order of Arm, Best Overall Response, and Duration on Study. (3) Use x-axis label of "Time Since T-cell Infusion (months)" and begin the axis (origin) at the start of lymphodepletion. (4) Remove all indication of diagnosis and prior therapies. (5) Show symbols or colored lines for: first confirmed response (star), SAE (asterisk), progression (diamond or other polygon), transfer to LTFU study (dot), ongoing participation in the study (blue line), date of first pembro (triangle), and ongoing status (at the time of analysis, arrow pointing to the right). (6) Show first date of progression, even if not confirmed. Please add a footnote to explain which subjects did not have confirmed progression. Not aligned w/study 208469 (MRCLS). | SAC | | | | |
| Safety: | Safety: Figures | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable | | | |
| 3.0640 | mITT | [Non-Standard]<br>SAFE_F1 | Plot of Prior Therapy Information by Treatment Arm | (1) Show all subjects on the same plot; do not show by treatment arm. Instead, add Arm label as an additional column to the right of Age/Sex. (2) Sort the Subject ID (y-axis) in ascending order of Arm, Best Overall Response, and Duration on Study. (3) Use x-axis label of "Time Since Tcell Infusion (months)". Begin the axis (origin) at the earliest diagnosis date (i.e., make sure the axis is expansive enough to show all diagnosis dates). End the axis at point of T-cell infusion. (4) Show symbols or colored lines for: Diagnosis, SAE, Leukapheresis, Surgery, Radiotherapy, Stem Cell Therapy (note that stem cell therapy + conditioning chemo represent a single regimen), Systemic Therapy Regimen 1, Regimen 2, Regimen 3, etc., and Lymphodepleting Chemotherapy. (5) Consider imputation of prior therapy dates in order to show duration on therapy. Add footnote: "Note: Start and end dates of prior therapy are imputed for missing day.' Not aligned w/study 208469 (MRCLS). | SAC | | | |

| Safety: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Labora | tory | | | | |
| 3.0650 | mITT | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin – eDISH | IDSL Include both treatment arms on same plot (same axes), with arms differentiated by color or pattern. Align w/study 208469 (MRCLS). | SAC |
| 3.0660 | mITT | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT | IDSL Include both treatment arms on same plot (same axes), with arms differentiated by color or pattern. Align w/study 208469 (MRCLS). | SAC |
| 3.0670 | mITT | [Non-Standard]<br>SAFE_F3 | Plot of Hematology Data Over Time | Produce a separate plot for neutrophils, lymphocytes, platelets, and hemoglobin (page-by lab test) Legend should list subjects by treatment arm, but subjects should not be grouped by treatment arm in the figure (each subject should have a unique color) X-axis units should be days starting at day -14.and ending at day 90. Not aligned w/study 208469 (MRCLS) | SAC |

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| ECG | | | | | |
| 3.0680 | mlTT | OECG4 | QTc Shifts from Baseline to Worst-Case Post Baseline | IDSL Include both treatment arms in same plot (same axes), with arms differentiated by color or pattern. Create separate plots for the 2 QTc correction methods (QTcB vs. QTcF). Align w/study 208469 (MRCLS). | SAC |

208470

## 14.12.9. Biomarkers Tables

| Biomar | Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Anti-N | Y-ESO-1 Antibo | odies | | | |
| 3.0690 | mITT | [Non-Standard]<br>BIO_T1 | Summary of Anti-NY-ESO-1 TCR(c259) Antibodies (ATA) | Align w/study 208469 (MRCLS). Only if data are available | SAC |

208470

## 14.12.10. Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Persist | ence of NY-ES | O-1 <sup>c259</sup> T | | | |
| 4.0010 | mITT | [Non-<br>Standard]<br>PK_T1 | Summary of Derived Persistence Parameters | Only report peak expansion (i.e. not by scheduled visits). Report overall and by responders vs. non-responders. Add total "by group" page. Display by type of persistence if BMMC data is available. Add footnote: "Note: Samples collected within 4 days of day 28 are treated as day 28 when calculating AUC(0-28)" Not aligned w/study 208469 (MRCLS). | SAC |
| 4.0020 | mITT | [Non-<br>Standard]<br>PK_T2 | Summary of Log-Transformed Derived Persistence Parameters | Report overall and by responders vs. non-responders. Add total "by group" page. Display by type of persistence if BMMC data is available. Add footnote: "Note: Samples collected within 4 days of day 28 are treated as day 28 when calculating AUC(0-28)" Not aligned w/study 208469 (MRCLS). | SAC |

208470

# 14.12.11. Pharmacokinetic Figures

| Pharmaco | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Persisten | ce of NY-ESO-19 | <sup>2259</sup> T | | | |
| 4.0030 | mITT | [Non-Standard]<br>PK_F2 | Distribution of Peak Expansion | Updated to dot plot. Please show both treatment arms on the same plot, with different colors for each arm. Plot by responders vs. non-responders. Page by type of persistence if BMMC data is available. Not aligned w/study 208469 (MRCLS). | SAC |
| 4.0040 | mITT | [Non-Standard]<br>PK_F1 | Persistence Profile by Subject | Plot by treatment arm. Present with x-axis sufficient to see all follow-up. Add subject numbers into the legend, add symbols at analysis timepoints, and differentiate subjects with symbols and tine types X-axis and Y-axis should be same for each treatment arm. Label X-axis "Study Day" rather than "Time from T-cell Infusion (Days)". Not aligned w/study 208469 (MRCLS). | SAC |
| 4.0050 | mITT | [Non-Standard]<br>PK_F1 | BMMC Persistence Profile by Subject | Present with x-axis sufficient to see all follow-up. Not aligned w/study 208469 (MRCLS). | SAC |

208470

# 14.12.12. ICH Listings

| ICH: Listi | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Subject D | isposition | | | | |
| 0010 | Screened | ES7 | Listing of Reasons for Screen Failure | Only include subjects that were screen failures; do not include "Run-In" elements or optional column "Type of Failure" Note that rescreened subjects that screen fail twice will appear twice in listing. Report as captured on CRF | SAC |
| 0020 | ITT | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 Do not include columns "Reason Term(s)", "Was a follow-up phone contact attempted 3 times?" & " Was a follow-up certified letter mailed?" from GSK standard mock as not collected in this study. Align w/study 208469 (MRCLS). | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 0030 | ITT | [Non-Standard]<br>POP_L5 | Listing of Study Treatment Status | ICH E3 Present this listing by treatment arm. Please include: Leukapheresis date, Lymphodepletion, T Cell Infusion Date, Time between Leukapheresis and T Cell Infusion, Transduced Dose, Completed Treatment Phase, Date of Discontinuation/Completion of Treatment Phase/Duration on Study (days), Reason for Discontinuation/Completion of Treatment Phase, End of Study Status Reason, and Death Date. Please insert a footnote: "Duration on Study refers to duration of follow-up on treatment phase." Not aligned w/study 208469 (MRCLS). | SAC |
| 0040 | mITT | ODMOD12A | Listing of Dose Delays (Pembrolizumab) | Do not include 'Primary reason for Delay/Specify' column Insert footnote: "Note: Duration of Delays = actual start date of current dose – expected start date of dose. Expected start date of dose=actual start date of previous dose + 21." Not aligned w/study 208469 (MRCLS) | SAC |
| 0050 | mITT | SD2 | Listing of Reasons for Study Treatment Discontinuation (Pembrolizumab) | ICH E3 Arm 2 only Not aligned w/study 208469 (MRCLS). | SAC |

| ICH: Listi | ings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Population | ons Analysed | | | | 1 |
| 0060 | Screened | SP3 | Listing of Subjects Excluded from Any Population | ICH E3 Include all subjects in population for display. Include columns to indicate exclusion ('Y') from Enrolled, ITT, and mITT populations. Drop "Date of Deviation/ Study day" and "Category/Coded Term" columns. Populate "Criteria" column with reason for exclusion from first: "SUBJECT NOT ELIGIBLE FOR APHERESIS", "SUBJECT NOT APHERESED", "SUBJECT NOT INFUSED". Align w/study 208469 (MRCLS). | SAC |
| Protocol | Deviations | | | | |
| 0070 | ITT | DV2 | Listing of Important Protocol Deviations | ICH E3<br>Align w/study 208469 (MRCLS). | SAC |
| 0800 | ITT | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3<br>Align w/study 208469 (MRCLS). | SAC |
| Demogra | phic and Basel | ine Characteristics | | | |
| 0090 | ITT | DM2 | Listing of Demographic Characteristics | ICH E3 Present this listing by treatment arm. Add BMI, BSA, and Race. Align w/study 208469 (MRCLS). | SAC |
| Prior and | Concomitant N | Medications | | | |
| 0100 | ITT | BP4 | Listing of Blood Products | Include all blood products. Align w/study 208469 (MRCLS). | SAC |

| ICH: Listi | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 0110 | ITT | CM3 | Listing of Medications | IDSL Include all collected medications, do not subset on concomitant medication study phase Replace "Started Pre-Trial" column with "Prior / Concomitant" (identified per Appendix 4) | SAC |
| Exposure | ) | | | | |
| 0120 | ITT | [Non-Standard]<br>POP_L3 | Listing of Leukapheresis, Lymphodepletion, T-cell, and Pembrolizumab Infusion Dates | ICH E3 With the exception of Pembro being added, this listing should align w/study 208469 (MRCLS). | SAC |
| 0130 | ITT | [Non-Standard]<br>POP_L1 | Listing of Exposure to Lymphodepletion Chemotherapy | ICH E3 One column for Fludarabine dose Align w/study 208469 (MRCLS). As per MRCLS, please remove MESNA. | SAC |
| 0140 | ITT | [Non-Standard]<br>POP_L2 | Listing of Exposure to T-cell Infusion | ICH E3<br>Align w/study 208469 (MRCLS). | SAC |
| 0150 | ITT | OEX8B | Listing of Exposure to Pembrolizumab | ICH E3 For subjects in Arm 2 only. Replace Cycle with Visit. Not aligned w/study 208469 (MRCLS). | SAC |

| ICH: Listin | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Adverse E | ents | | | | • |
| 0160 | ITT | AE8 | Listing of All Adverse Events | ICH E3 Present this listing by treatment arm. Report time from first T-cell Infusion. Use "Time Since T-cell Infusion" instead of Time Since First Dose/Time Since Last Dose. Add MM Combo specific "action taken" column. With the exception of the added "action taken" (specific to MM Combo), this listing should align w/study 208469 (MRCLS). | SAC |
| 0170 | ITT | AE8 | Listing of Adverse Events Leading to Dose Interruption, Dose Reduction, or Permanent Discontinuation of Pembrolizumab | For subjects in Arm 2 only. Not aligned w/study 208469 (MRCLS). | SAC |
| 0180 | ITT | [Non-Standard]<br>SAFE_L1 | Listing of Delayed Adverse Events | ICH E3 Report time from first T-cell Infusion. Use "Time Since T-cell Infusion" instead of Time Since First Dose/Time Since Last Dose. | SAC |
| 0190 | ITT | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 All AEs. Align w/study 208469 (MRCLS). | SAC |
| 0200 | ITT | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL<br>Align w/study 208469 (MRCLS). | SAC |

| ICH: List | ings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Adverse | Events of Spec | ial Interest | | | <del>'</del> |
| 0210 | mITT | [Non-Standard]<br>SAFE_L1 | Listing of AESI (Focused List) | Use Focused Scope List. Sort by USUBJID, AEDECOD, ASTDT, AENDT. Present by treatment arm and by AESI. Align w/study 208469 (MRCLS). | SAC |
| 0220 | mITT | [Non-Standard]<br>SAFE_L1 | Listing of Haematopoietic Cytopenias (Comprehensive List) | Use Comprehensive Scope List. Sort by USUBJID, AEDECOD, ASTDT, AENDT. Present by treatment arm. Align w/study 208469 (MRCLS). | SAC |
| 0225 | mITT | [Non-Standard]<br>SAFE_L6 | Listing of CARTOX and ICE Score | Align w/study 208469 (MRCLS) | SAC |
| Serious | and Other Signi | ficant Adverse Events | | | |
| 0230 | ITT | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3<br>Align w/study 208469 (MRCLS). | SAC |
| 0240 | ITT | AE14 | Listing of Reasons for Considering as a Serious<br>Adverse Event | ICH E3 Add PAN12. Align w/study 208469 (MRCLS). | SAC |
| 0250 | ITT | PAN12 | Listing of COVID-19 Assessments and Symptom<br>Assessments for Subjects with COVID-19 Adverse<br>Events | If data exists | SAC |
| Death | | | | | |
| 0260 | ITT | DD3 | Death Profile | Align w/study 208469 (MRCLS). | SAC |

| ICH: Listi | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Hepatobiliary (Liver) | | | | | |
| 0270 | ITT | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | IDSL Update columns "Time Since First / Last Dose (days)" of LIVER5 mock with "Time Since First T-cell Infusion" & "Time Since Last T-cell Infusion". Align w/study 208469 (MRCLS). | SAC |
| 0280 | ІТТ | LIVER15 | Liver Stopping Event Profile | IDSL Update variables "Time Since First / Last Dose (days)" of LIVER15 mock with "Time Since First T-cell Infusion" & "Time Since Last T-cell Infusion". Align w/study 208469 (MRCLS). | SAC |
| 0290 | ІТТ | LIVER13 | Listing of Subjects Meeting Hepatobiliary Laboratory<br>Criteria Post-Baseline | IDSL Please make sure this is derived correctly by considering all liver function criteria specified in the LIVER IDSL doc. Align w/study 208469 (MRCLS). | SAC |
| All Labora | atory | | | | |
| 0300 | ІТТ | LB5A | Listing of All Laboratory Data | ICH E3 Combining all laboratory data (chem, hem, etc.) in one listing, including biomarker data but NOT including urinalysis data. Align w/study 208469 (MRCLS). | SAC |
| 0310 | ITT | UR2A | Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | ICH E3<br>Align w/study 208469 (MRCLS). | SAC |

| ICH: List | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Replicati | Replication Competent Lentivirus (RCL) | | | | |
| 0320 | mITT | LB5A | Listing of VSV-G DNA (RCL) Data | Align w/study 208469 (MRCLS). | SAC |
| 0330 | mITT | [Non-Standard]<br>SAFE_L2 | Listing of Integration Site Analysis Results | This is a supplemental display to the table summary "Summary of Subjects Showing Monoclonality of Genetically Modified T-cell Population" (which uses SAFE_T3). Create only if data are available. Align w/study 208469 (MRCLS). | SAC |
| Pharmac | okinetic | | | | |
| 0340 | mlTT | [Non-Standard]<br>PK_L1 | Listing of Persistence Data | Present this listing by treatment arm. Present by persistence type if BMMC data are available. Show time to loss of 25%, 50% and 75% of peak expansion, peak expansion, time to peak expansion, and AUC(0-28). With the exception of the added AUC(0-28) parameter, this listing should align w/study 208469 (MRCLS). | SAC |
| Biomark | ers | | | | |
| 0350 | mITT | [Non-Standard]<br>BIO_L1 | Listing of Anti-NY-ESO-1 Antibodies | Align w/study 208469 (MRCLS). Only if data are available | SAC |

| ICH: Listi | ngs | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| ECG | ECG | | | | |
| 0360 | ITT | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | IDSL Update PCI footnote to use oncology definition "Clinical Importance is defined as Grade 2 or Higher (QTc>480), or QTc increase of >30 msec" (as in OECG5A). Align w/study 208469 (MRCLS). | SAC |
| 0370 | ITT | EG5 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding | IDSL "Clinically significant change from baseline" and "Clinically Significant Abnormality" in this standard shell are not collected in this study so cannot be reported – drop from display. | SAC |
| V'(-1.0' | | | | Align w/study 208469 (MRCLS). | |
| Vital Sign | ITT | OVT7A | Listing of Vital Signs with Values of Potential Clinical Importance | IDSL<br>Align w/study 208469 (MRCLS). | SAC |
| Response | е | | | | |
| 0390 | ITT | [Non-Standard]<br>EFF_L2 | Listing of Investigator-Assessed Responses (with confirmation) (IMWG 2016) | Present this listing by treatment arm. Please ensure that an additional column is included to display "by-visit" Confirmed Response, to the right of the column of "by-visit" responses. Not aligned w/study 208469 (MRCLS). | SAC |

| ICH: Listi | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Time to Event | | | | | |
| 0400 | mITT | TTE9 | Listing of Investigator-Assessed Time to Response (IMWG 2016) | Use T-cell infusion date. Include optional "New Anti-Cancer Therapy Start Date" column. Align w/study 208469 (MRCLS). | SAC |
| 0410 | mITT | TTE9 | Listing of Investigator-Assessed Duration of Response (IMWG 2016) | Present this listing by treatment arm. Add Initial Confirmed Response. Use T-cell infusion date. Include optional "New Anti-Cancer Therapy Start Date" column. Include footnote: "Note: Duration of Response is defined as the interval between the initial date of the confirmed response (sCR, CR, VGPR, or PR) and the date of confirmed progressive disease or death among subjects with a confirmed response per IMWG 2016." Align w/study 208469 (MRCLS). | SAC |
| 0420 | mITT | TTE9 | Listing of Investigator-Assessed Progression Free Survival (IMWG 2016) | Present this listing by treatment arm. Use T-cell infusion date Include optional "New Anti-Cancer Therapy Start Date" column. Similar to the footnote used in the DoR listing above, add a footnote that defines PFS as including confirmed progressive disease. Align w/study 208469 (MRCLS). | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 0430 | mITT | TTE9 | Listing of Overall Survival | Use T-cell infusion date. Exclude optional "New Anti-Cancer Therapy Start Date" column. Align w/study 208469 (MRCLS). | SAC |

208470

# 14.12.13. Non-ICH Listings

| Non-ICH: | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Disease | Characteristic | s | | | |
| 0440 | ITT | DC3 | Listing of Disease Characteristics at Initial Diagnosis | Present this listing by treatment arm. Please report: date of initial diagnosis, time from initial diagnosis to screening ICF signed (in months), stage at diagnosis, histologic type, % clonal bone marrow plasma cells, presence and type of end organ damage, presence and type of plasmacytoma, and chromosomal aberrations. Remove primary neoplasm type under study and study specific category (as they are not relevant) and remove histologic grade (as it is not collected). Not aligned w/study 208469 (MRCLS). | SAC |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 0450 | ITT | [Non-Standard]<br>POP_L4 | Listing of Disease Characteristics at Screening | Present this listing by treatment arm. Please report: type of multiple myeloma, HLA status (date, allele 1, allele 2), NY-ESO-1 biopsy date and status, LAGE-1a (date, status), number of systemic therapy / radiotherapy regimens prior to leukapheresis, and receipt of stem cell transplant/therapy prior to leukapheresis (Y/N) for each of 2 subtypes (autologous vs. allogeneic). Also, use the new derivation of lines of systemic therapy (i.e., count systemic therapy + conditioning chemo associated w/stem cell therapy) – please add a footnote that makes this clear. Not aligned w/study 208469 (MRCLS). | SAC |

| Non-ICH: Listings | | | | |
|---|---|---|---|---|
| Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| ncer Therapies | | | | |
| IΠ | AC6 | Listing of Prior Systemic Anti-Cancer Therapy | Present this listing by treatment arm. In addition to the Most Recent Response, please include "Best Response" in the same column (to be shown first) and "MRD" (to be shown last). Remove "Reason for Stopping" (as not collected for prior systemic therapy) and replace it with "Disease Refractory to Regimen (Y/N)". Add "Intent" (i.e., treatment intent). Add final column with header of "Started after Leukapheresis?/Bridging Therapy?" "Note: This listing includes all systemic therapy prior to lymphodepletion." Sort by regimen. Conditioning chemotherapies (associated with stem cell therapy) and stem cell therapy should appear in this listing Not aligned w/study 208469 (MRCLS). | SAC |
| | Population | Population IDSL / Example Shell | Population IDSL / Example Shell Title | Programming Notes |

| Non-ICH | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 0470 | ITT | AC7 | Listing of Anti-Cancer Radiotherapy | List all radiotherapy before lymphodepletion and flag the ones occurring between leukapheresis and lymphodepletion as "Started after Leukapheresis". Use T-cell infusion date. Include optional "New Anti-Cancer Therapy Start Date" column. Add final column with header of "Transition Therapy" Add footnotes: "Note: This listing includes all radiotherapy received by the subject." "Note: Transition therapies include all therapy received after leukapheresis and before lymphodepletion." Align w/study 208469 (MRCLS). | SAC |
| 0480 | ІТТ | FAC3 | Listing of On-Study Anti-Cancer Therapy | Include "Time to Progression (Days)" but not "Overall Survival (Days)". Use date of "first progression" even if not confirmed for TTP column. Footnote any subject with unconfirmed PD. Includes radiotherapy, systemic therapy, and stem cell therapy Align w/ study 208469 (MRCLS) | SAC |

| Non-ICH | : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Symptor | Symptoms, Concomitant Medications and Procedures Related to Adverse Events of Special Interest | | | | |
| 0490 | ІТТ | [Non-Standard]<br>SAFE_L4 | Listing of Symptoms, Concomitant Medications, and Procedures Related to Cytokine Release Syndrome (CRS) | Present this listing by treatment arm. Add column showing list of all symptoms. Align w/study 208469 (MRCLS). | SAC |
| 0500 | ITT | [Non-Standard]<br>SAFE_L5 | Listing of Symptoms, Concomitant Medications, and Procedures Related to Graft versus Host Disease (GvHD) | Present this listing by treatment arm. Add column showing list of all symptoms. Align w/study 208469 (MRCLS). | SAC |
| Surgical | Procedures | | | | |
| 0510 | ITT | OSP3 | Listing of Prior Cancer-Related Surgical Procedures | List all surgeries before lymphodepletion and flag the ones occurring between leukapheresis and lymphodepletion as "Started after Leukapheresis?" List Surgery Intent and Site and Date of Surgery. Add footnote: "Note: This listing includes all cancer-related surgeries prior to T-cell | SAC |
| 0520 | ITT | ITT OSP3 | Listing of On-Study Cancer-Related Surgical Procedures | infusion." Align w/study 208469 (MRCLS). List Site and Date of Surgery. Align w/study 208469 (MRCLS). | SAC |

208470

## 14.13. Appendix 13: Example Mock Shells for Data Displays

Data Display Specification will be made available on request

#### 208470

# 14.14. Appendix 14: Combined Preferred Terms

| Combined Term | MedDRA Preferred term | PT Code | |
|---|---|---|---|
| Anemia/RBC decreased | Anemia | 10002034 | PT |
| Cytokine Release Syndrome (CRS) | Cytokine Release Syndrome | 10052015 | PT |
| | Cytokine Storm | 10050685 | PT |
| Acute GVHD - Skin | Acute graft versus host disease in skin | 10066262 | PT |
| Acute GVHD - Gut (Liver and Intestine) | Acute graft versus host disease in liver | 10066263 | PT |
| | Acute graft versus host disease in intestine | 10066264 | PT |
| Acute GVHD - Other (Lung, Bone Marrow, not specified) | Acute graft versus host disease | 10066260 | PT |
| Chronic GVHD - Skin | Chronic graft versus host disease in skin | 10072159 | PT |
| Chronic GVHD - Gut (Liver and Intestine) | Chronic graft versus host disease in liver | 10072160 | PT |
| | Chronic graft versus host disease in intestine | 10072158 | PT |
| Chronic GVHD Other - (Lung, Bone Marrow, not specified) | Chronic graft versus host disease | 10066261 | PT |
| Unspecified GVHD - Skin | Graft versus host disease in skin | 10064675 | PT |
| Unspecified GVHD - Gut (Liver and Intestine) | Graft versus host disease in liver | 10064676 | PT |
| | Graft versus host disease in gastrointestinal tract | 10075160 | PT |
| Unspecified GVHD - Other (Lung, Bone Marrow, not specified) | Graft versus host disease | 10018651 | PT |
| | Graft versus host disease in eye | 10074563 | PT |
| | Graft versus host disease in lung | 10067742 | PT |
| | Prophylaxis against graft versus host disease | 10053239 | PT |

| Combined Term | MedDRA Preferred term | PT Code | |
|---|---|---|---|
| | Transfusion associated graft versus host | | |
| | disease | 10070895 | PT |
| | Engraftment syndrome | 10050684 | PT |
| Leukopenia/WBC decreased | White blood cell count decreased | 10047942 | PT |
| | Leukopenia | 10024384 | PT |
| Lymphopenia/Lymphocyte count decreased | Lymphocyte count decreased | 10025256 | PT |
| | CD4 lymphocytes decreased | 10007839 | PT |
| | CD8 lymphocytes decreased | 10056283 | PT |
| Neutropenia/Neutrophil count decreased | Neutrophil count decreased | 10029366 | PT |
| | Neutropenia | 10029354 | PT |
| Rash/Rash maculo-papular | Rash maculo-papular | 10037868 | PT |
| • | Rash | 10037844 | PT |
| | Rash erythematous | 10037855 | PT |
| Thrombocytopenia/Platelet count decreased | Platelet count decreased | 10035528 | PT |
| | Thrombocytopenia | 10043554 | PT |
| | MedDRA version 21.1 for PT codes | | |

208470

#### 14.15. Appendix 15: Adverse Event Collapsing Rules

#### 1. Collapsing AE Segments with a Common AE Preferred Term (PT) into Unique Events based on the Start and End Dates

For each unique subject, the AE records (segments) with the same AE preferred term will be collapsed into one unique AE event based on the start and end dates below.

#### 1.1. Multiple AE Segments with Overlapped or Continuous Start/End Dates

Multiple AE segments with a common preferred term (PT, variable=ADAE.AEDECOD) that occurred around the same time; defined as:

If a segment starts no more than one day (i.e.,  $\leq 1$  day) prior, on, or after the previous segment's end date, it is considered as an 'event'.

If the gap between the start date of a segment and the end date of previous segment is greater than one complete day (i.e., > 1 day), then consider these segments as different events.

If partial start or end dates for any AE segments, then consider these segments as separate events.

#### \*\*\* NOTE: Handling of partial dates or completely missing dates

Partial dates or completely missing dates will not be imputed.

The reason for not using imputed dates is due to the small number of partial / or completely missing dates. Furthermore, using imputed dates might create additional error of up to 30 days off for the AE start or AE end dates, and can be up to 60 days off for the duration of AE.

208470

#### 1.2.Sort Adverse Events (AE)

For any AE event identified above:

Sort the AEs segments by study ID (ADAE.STUDYID), unique subject ID (ADAE.USUBJID), AE preferred term (ADAE.AEDECOD), AE start date (ADAE.AESTDTC), and AE end date (ADAE.AEENDTC). The sorting will include all AE segments with complete or partial start / end dates.

#### 1.3. Create Derived Variables in ADAE ADaM SAS Dataset

Based on the ADAE dataset sorted above under Section 1.2, for each unique subject, create the following derived variables in the ADAE ADaM SAS dataset:

#### 1) ANL01FL: Flag for the unique AE

a) Collapsed AE Segments

For collapsed AE segments. based on the ADAE dataset sorted above under Section 1.2:

- derive the flag variable: <u>ANL01FL="Y" on the first record for each collapsed AE (i.e. the earliest segment within each collapsed AE with the same ADAE.AEDECOD)</u>. In case if the AE segment of the collapsed AEs started before Lymphodepletion and ending after it, then populate the ANL01FL='Y' on very first Treatment emergent record. If there is only one record (segment) which started before lymphodepletion and ended after lymphodepletion then populate ANL01FL='Y' on that record only.
- Otherwise ANL01FL="" (Missing).
- b) AE Events Comprised of a Single Row (No Collapsing Needed)
  - derive the flag variable: ANL01FL="Y" for each single segment AE event.

#### 2) EVTSEQ: Sequence number of each unique AE with the same PT

Create a sequence number, EVTSEQ, for each unique AE within the same ADAE.AEDECOD.

For each unique subject within each unique AE preferred term, this variable will be recorded as <u>the sequential</u> <u>number to identify all unique adverse events (including both single segment events (i.e., no collapsing needed) and collapsed events from multiple segments) based on the sorting order chronologically addressed above under Section 1.2.</u>

#### a) Collapsed AE Segments

Each collapsed AE and its corresponding composed segments will have the same sequence numbers (i.e., if multiple segments/records are qualified for being collapsed into one unique AE (i.e., all those records will have same value for the derived variable EVTSEQ for that corresponding subject within the same collapsed AE).

#### b) Single Segment AE Records

Each single segment AE event (i.e., un-collapsed event) will have different unique sequence number separately

#### c) AE Segments with partial start or end dates

Each AE segment with partial start or end dates will have different unique sequence number starting from 99XXX, where XXX=001, 002, ...

#### \* NOTE:

For those subjects who received 2 T-cell infusions, the sequential number will be based on both infusion periods combined (i.e., the assigned sequential number will be independent of T-cell infusion periods).